CLINICAL TRIAL: NCT00442546
Title: A Multicenter, Double-Blind Randomized, Placebo-Controlled Study Of The Efficacy And Safety Of Pregabalin In The Treatment Of Subjects With Post-Operative Pain Following Total Knee Arthroplasty (TKA)
Brief Title: Efficacy And Safety Of Pregabalin For Pain Following Total Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081133
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis; Postoperative Pain
Keywords: opioid
MeSH Terms: conditions — Osteoarthritis; Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: pregabalin
- 2 (Experimental)
  Interventions: Drug: pregabalin
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin — 150 milligram (mg)/ day (double blind)
  Arms: 1
Drug: pregabalin — 300 mg/day (double blind)
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
Pregabalin added to the standard of care with dosing starting preoperatively and continuing for up to 6 weeks post surgery will decrease the intensity of post-operative pain following total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with osteoarthritis (OA) undergoing elective TKA under regional anesthesia (neuroaxial with or without peripheral nerve block).
* Subjects able to demonstrate sufficient psychomotor dexterity and cognitive capacity to use Patient Controlled Analgesia/Patient Controlled Epidural Analgesia if used as part of the standard of care.
* The subject's preoperative health is graded as American Society of Anesthesiology Class 1 to Class 3

Exclusion Criteria:

* Subjects undergoing revision, unicompartmental, bilateral total knee arthroplasty or subjects with planned second knee total knee arthroplasty at time of present procedure.
* Subjects with inflammatory arthritides (i.e., rheumatoid arthritis, lupus, ankylosing spondylitis, psoriatic arthritis); Lyme disease.
* Subjects with fibromyalgia and or other chronic pain syndromes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (24):
  - Pfizer Investigational Site, Northport, Alabama
  - Pfizer Investigational Site, Tuscaloosa, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Galesburg, Illinois
  - Pfizer Investigational Site, Lafayette, Louisiana
  - Pfizer Investigational Site, New Iberia, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Egg Harbor, New Jersey
  - Pfizer Investigational Site, Pomona, New Jersey
  - Pfizer Investigational Site, Voorhees Township, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Upper Arlington, Ohio
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, King of Prussia, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- [Derived] Singla NK, Chelly JE, Lionberger DR, Gimbel J, Sanin L, Sporn J, Yang R, Cheung R, Knapp L, Parsons B. Pregabalin for the treatment of postoperative pain: results from three controlled trials using different surgical models. J Pain Res. 2014 Dec 23;8:9-20. doi: 10.2147/JPR.S67841. eCollection 2015. PMID 25565885

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin (150 Milligrams [mg]): Pregabalin capsules orally 75 mg the evening before surgery (approximately 12 hours prior to surgery) followed by 75 mg approximately 2 hours before surgery followed by 150 mg/day (75 mg twice daily) for up to 6 post-operative weeks starting on Post-Operative Day 1 (POD 1).
- Pregabalin (300 mg): Pregabalin capsules orally 150 mg the night before surgery (approximately 12 hours prior to surgery) followed by 150 mg approximately 2 hours before surgery followed by 300 mg/day (150 mg twice daily) for up to 6 post-operative weeks starting on POD 1.
- Placebo: Matching Placebo capsules orally: 1 dose the evening before surgery (approximately 12 hours prior to surgery), 1 dose approximately 2 hours before surgery followed by twice daily dosing for up to 6 post-operative weeks starting on POD 1.
Period: Overall Study
Arm/Group | Pregabalin (150 Milligrams [mg]) | Pregabalin (300 mg) | Placebo
Started | 103 | 100 | 104
Received Treatment | 98 | 96 | 98
Completed | 77 | 63 | 71
Not Completed | 26 | 37 | 33
Not completed — Adverse Event | 11 | 17 | 13
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Other | 4 | 9 | 6
Not completed — Withdrawal by Subject | 5 | 5 | 7
Not completed — Randomized But Not Treated | 5 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin (150 mg): Pregabalin capsules orally 75 mg the evening before surgery (approximately 12 hours prior to surgery) followed by 75 mg approximately 2 hours before surgery followed by 150 mg/day (75 mg twice daily) for up to 6 post-operative weeks starting on POD 1.
- Total: Total of all reporting groups
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo | Total
Number analyzed (Participants) | 98 | 96 | 98 | 292
Age, Customized [Number; unit: participants]
  18 to 44 years | 1 | 2 | 4 | 7
  45 to 64 years | 52 | 44 | 49 | 145
  > = 65 years | 45 | 50 | 45 | 140
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 61 | 54 | 175
  Male | 38 | 35 | 44 | 117

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Worst Pain Score in Daily Diaries Using the Worst Pain Item of the Modified Brief Pain Inventory - Short Form (m-BPI-sf)
Description: The mBPI-SF is a self administered questionnaire developed to assess pain severity and pain interference with functional activities during a 24-hour period prior to evaluation. For the Worst Pain item of the m-BPI-sf scale (11 point Likert scale; range: 0 [no pain] to 10 [pain as bad as you can imagine]), subjects were asked to rate their pain by marking an "X" in one of the ten boxes that best described their pain at its worst in the last 24 hours post surgery and at least 12 hours after discontinuation of the peripheral nerve block or neuroaxial block.
Time Frame: 48 hours after surgery
Population: Modified Intent-to-Treat (MITT) Population=all ITT subjects who took 12 and 2 hours pre-surgery study medications, had no surgical or anesthetic complications during total knee replacement surgery and had at least 1 post surgery primary efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 78 | 82 | 75
scores on a scale | 7.041 (0.267) | 6.740 (0.264) | 7.079 (0.279)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Test type: Superiority or Other; p = 0.9185, ANOVA — A step-down procedure was used for multiple comparisons adjustment. If the difference between the high dose and placebo groups was statistically significant (p<0.05), then the next step conducted where the low dose group was compared to placebo; Least squares means from the analysis of variance (ANOVA) model with main effects of treatment and center and Baseline mean worst pain score; Mean Difference (Final Values) = -0.038, 95% CI [-0.766 to 0.691], Standard Error of Mean 0.370 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Test type: Superiority or Other; p = 0.3619, ANOVA — [p-value comment as in outcome 1, analysis 1]; Least squares means from the ANOVA model with main effects of treatment and center and Baseline mean worst pain score; Mean Difference (Final Values) = -0.339, 95% CI [-1.070 to 0.392], Standard Error of Mean 0.371 — Mean difference (final values) = Least squares mean difference

2. Secondary Outcome: Cumulative Total Amount of Opioids Used During the Entire Hospital Stay
Description: Total cumulative dose calculated as mg of oral morphine equivalent and included opioids given by any route (patient controlled analgesia [PCA] pump, parenteral bolus or oral). Results for daily total not including pregabalin (not an opioid). Statistical model included main effect of treatment group and center. 1 subject at 144 h, 300 mg=non-missing data. Due to small sample size (N=1, 300 mg; N=5, other groups) and large opioid consumption for another subject in same center, least squares mean (300 mg, 144 h) is negative.
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours, 168 hours, 192 hours, 216 hours
Population: MITT. There were not enough subjects with data at 168, 192, and 216 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: mg of oral morphine equivalent
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 85 | 86 | 84
mg of oral morphine equivalent
  24 hours (n=85, 86, 84) | 151.790 (14.210) | 152.306 (14.313) | 167.854 (14.573)
  48 hours (n=82, 81, 83) | 86.402 (12.057) | 93.846 (12.292) | 122.830 (12.304)
  72 hours (n=60, 60, 60) | 55.654 (9.175) | 48.713 (9.420) | 52.895 (9.851)
  96 hours (n=32, 39, 35) | 31.976 (7.928) | 24.758 (7.861) | 35.332 (8.354)
  120 hours (n=12, 6, 13) | 27.520 (13.146) | 14.235 (17.684) | 27.559 (13.306)
  144 hours (n=5, 1, 5) | 33.956 (12.019) | -64.544 (28.633) | 73.956 (16.720)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.4091, ANOVA; Mean Difference (Final Values) = -16.065, 95% CI [-54.332 to 22.203], Standard Error of Mean 19.426 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.4234, ANOVA; Mean Difference (Final Values) = -15.548, 95% CI [-53.740 to 22.645], Standard Error of Mean 19.388 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.0284, ANOVA; Mean Difference (Final Values) = -36.428, 95% CI [-68.972 to -3.884], Standard Error of Mean 16.517 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.0816, ANOVA; Mean Difference (Final Values) = -28.985, 95% CI [-61.632 to 3.663], Standard Error of Mean 16.570 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.8147, ANOVA; Mean Difference (Final Values) = 2.759, 95% CI [-20.446 to 25.964], Standard Error of Mean 11.752 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.7187, ANOVA; Mean Difference (Final Values) = -4.182, 95% CI [-27.064 to 18.700], Standard Error of Mean 11.589 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.7416, ANOVA; Mean Difference (Final Values) = -3.356, 95% CI [-23.516 to 16.804], Standard Error of Mean 10.148 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.2577, ANOVA; Mean Difference (Final Values) = -10.574, 95% CI [-29.017 to 7.869], Standard Error of Mean 9.283 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.9982, ANOVA; Mean Difference (Final Values) = -0.039, 95% CI [-36.431 to 36.352], Standard Error of Mean 17.387 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.5552, ANOVA; Mean Difference (Final Values) = -13.325, 95% CI [-59.756 to 33.107], Standard Error of Mean 22.184 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; 144 hours; Test type: Superiority or Other; p = 0.2032, ANOVA; Mean Difference (Final Values) = -40.000, 95% CI [-118.463 to 38.463], Standard Error of Mean 24.655 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; 144 hours; Test type: Superiority or Other; p = 0.0348, ANOVA; Mean Difference (Final Values) = -138.500, 95% CI [-258.354 to -18.646], Standard Error of Mean 37.661 — Mean difference (final values) = Least squares mean difference

3. Secondary Outcome: Opioids Used Post Discharge
Description: The amount of opioid use was calculated as mg of oral morphine equivalent and included opioids administered by any route (PCA pump, parenteral bolus, or oral). Weeks 2, 4, and 6 total daily doses were calculated by adding the cumulative doses during the 2 week period prior to the visit and dividing them by the number of days in the period. This outcome measure does not include pregabalin as it is not an opioid.
Time Frame: Week 2, Week 4, Week 6/Early Termination (ET)
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: mg of oral morphine equivalent
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 41 | 40 | 36
mg of oral morphine equivalent
  Week 2 (n=41, 40, 36) | 30.255 (3.515) | 27.692 (3.534) | 26.119 (3.789)
  Week 4 (n=33, 33, 30) | 37.130 (4.975) | 37.507 (4.911) | 34.271 (5.274)
  Week 6/ET (n=24, 28, 22) | 38.686 (6.261) | 35.945 (5.888) | 35.036 (6.401)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.3602, ANOVA; Mean Difference (Final Values) = 4.136, 95% CI [-4.790 to 13.062], Standard Error of Mean 4.499 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7352, ANOVA; Mean Difference (Final Values) = 1.573, 95% CI [-7.626 to 10.771], Standard Error of Mean 4.637 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6435, ANOVA; Mean Difference (Final Values) = 2.860, 95% CI [-9.392 to 15.111], Standard Error of Mean 6.156 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6123, ANOVA; Mean Difference (Final Values) = 3.237, 95% CI [-9.422 to 15.895], Standard Error of Mean 6.361 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.6356, ANOVA; Mean Difference (Final Values) = 3.650, 95% CI [-11.683 to 18.984], Standard Error of Mean 7.663 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9070, ANOVA; Mean Difference (Final Values) = 0.909, 95% CI [-14.593 to 16.411], Standard Error of Mean 7.747 — Mean Difference (Final Values) = Least Squares Mean Difference

4. Secondary Outcome: Analgesics Used During the Hospital Stay (Acetylsalicylic Acid, Ketorolac, and Paracetamol)
Description: Total dose for in-hospital visits was the total dose for the day.
Time Frame: 24 hours, 48 hours, 72 hours
Population: MITT. There were not enough subjects with data to calculate least squares mean values at 24 and 48 hours for Acetylalicyclic Acid and 72 hours for Ketorolac.
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 22 | 25 | 17
mg
  Acetylsalicylic Acid, 72 hours (n=3, 1, 1) | 235.175 (61.531) | 1442.025 (117.823) | 1425.825 (117.823)
  Ketorolac, 24 hours, (n=1, 4, 3) | 32.961 (57.230) | 53.432 (28.615) | 27.189 (31.346)
  Ketorolac, 48 hours, (n=2, 8, 4) | 20.553 (7.971) | 21.863 (3.862) | 23.473 (5.520)
  Paracetamol, 24 hours (n=14, 20, 16) | 1311.246 (359.886) | 1363.086 (283.808) | 1380.481 (309.224)
  Paracetamol, 48 hours (n=22, 25, 17) | 1357.030 (371.095) | 1368.880 (339.509) | 1263.337 (443.695)
  Paracetamol, 72 hours (n=12, 13, 16) | 446.050 (445.588) | 877.916 (403.657) | 1128.355 (347.457)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Acetylsalicylic Acid, 72 hours; Test type: Superiority or Other; p = 0.0656, ANOVA; Mean Difference (Final Values) = -1190.650, 95% CI [-2754.304 to 373.004], Standard Error of Mean 123.062 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Acetylsalicylic Acid, 72 hours; Test type: Superiority or Other; p = 0.9277, ANOVA; Mean Difference (Final Values) = 16.200, 95% CI [-1789.352 to 1821.752], Standard Error of Mean 142.100 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Ketorolac, 24 hours; Test type: Superiority or Other; p = 0.9350, ANOVA; Mean Difference (Final Values) = 5.771, 95% CI [-263.972 to 275.515], Standard Error of Mean 62.692 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Ketorolac, 24 hours; Test type: Superiority or Other; p = 0.6139, ANOVA; Mean Difference (Final Values) = 26.243, 95% CI [-164.494 to 216.980], Standard Error of Mean 44.330 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Ketorolac, 48 hours; Test type: Superiority or Other; p = 0.7760, ANOVA; Mean Difference (Final Values) = -2.920, 95% CI [-25.451 to 19.611], Standard Error of Mean 9.960 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Ketorolac, 48 hours; Test type: Superiority or Other; p = 0.8190, ANOVA; Mean Difference (Final Values) = -1.610, 95% CI [-17.066 to 13.846], Standard Error of Mean 6.833 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Paracetamol, 24 hours; Test type: Superiority or Other; p = 0.8603, ANOVA; Mean Difference (Final Values) = -69.235, 95% CI [-861.171 to 722.700], Standard Error of Mean 390.483 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Paracetamol, 24 hours; Test type: Superiority or Other; p = 0.9642, ANOVA; Mean Difference (Final Values) = -17.395, 95% CI [-796.945 to 762.155], Standard Error of Mean 384.376 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Paracetamol, 48 hours; Test type: Superiority or Other; p = 0.8476, ANOVA; Mean Difference (Final Values) = 93.693, 95% CI [-880.865 to 1068.251], Standard Error of Mean 484.957 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Paracetamol, 48 hours; Test type: Superiority or Other; p = 0.8185, ANOVA; Mean Difference (Final Values) = 105.543, 95% CI [-813.584 to 1024.670], Standard Error of Mean 457.374 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Paracetamol, 72 hours; Test type: Superiority or Other; p = 0.1792, ANOVA; Mean Difference (Final Values) = -682.304, 95% CI [-1696.759 to 332.150], Standard Error of Mean 495.241 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Paracetamol, 72 hours; Test type: Superiority or Other; p = 0.6216, ANOVA; Mean Difference (Final Values) = -250.439, 95% CI [-1278.347 to 777.469], Standard Error of Mean 501.808 — Mean Difference (Final Values) = Least Squares Mean Difference

5. Secondary Outcome: Analgesics Used Post Discharge (Acetylsalicylic Acid [Week 2] and Paracetamol [Weeks 2, 4, and 6]
Description: Weeks 2, 4, and 6 total daily doses were calculated by adding the cumulative doses during the 2 week period prior to the visit and dividing them by the number of days in the period.
Time Frame: Week 2, Week 4, Week 6/ET
Population: MITT.
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 7 | 14 | 7
mg
  Acetylsalicylic Acid, Week 2 (n=6, 1, 2) | 498.613 (130.446) | 797.463 (361.189) | 992.613 (291.687)
  Paracetamol, Week 2 (n=7, 13, 7) | 603.496 (232.179) | 665.574 (164.777) | 630.787 (247.693)
  Paracetamol, Week 4 (n=5, 12, 6) | 792.434 (412.260) | 779.226 (260.034) | 593.498 (375.124)
  Paracetamol, Week 6/ET (n=6, 14, 5) | 1128.952 (290.993) | 1098.840 (223.948) | 1385.873 (334.859)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Acetylsalicylic Acid, Week 2; Test type: Superiority or Other; p = 0.1996, ANOVA; Mean Difference (Final Values) = -494.000, 95% CI [-1452.720 to 464.720], Standard Error of Mean 301.253 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Acetylsalicylic Acid, Week 2; Test type: Superiority or Other; p = 0.6335, ANOVA; Mean Difference (Final Values) = -195.150, 95% CI [-1369.338 to 979.038], Standard Error of Mean 368.958 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Paracetamol, Week 2; Test type: Superiority or Other; p = 0.9290, ANOVA; Mean Difference (Final Values) = -27.291, 95% CI [-657.992 to 603.410], Standard Error of Mean 302.355 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Paracetamol, Week 2; Test type: Superiority or Other; p = 0.8937, ANOVA; Mean Difference (Final Values) = 34.787, 95% CI [-501.241 to 570.815], Standard Error of Mean 256.969 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Paracetamol, Week 4; Test type: Superiority or Other; p = 0.6912, ANOVA; Mean Difference (Final Values) = 198.937, 95% CI [-847.930 to 1245.804], Standard Error of Mean 491.153 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Paracetamol, Week 4; Test type: Superiority or Other; p = 0.6024, ANOVA; Mean Difference (Final Values) = 185.728, 95% CI [-558.248 to 929.704], Standard Error of Mean 349.047 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Paracetamol, Week 6/ET; Test type: Superiority or Other; p = 0.5372, ANOVA; Mean Difference (Final Values) = -256.921, 95% CI [-1120.551 to 606.709], Standard Error of Mean 407.391 — Mean Difference (Final Values) = Least Squares Mean Difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Paracetamol, Week 6/ET; Test type: Superiority or Other; p = 0.3948, ANOVA; Mean Difference (Final Values) = -287.032, 95% CI [-982.843 to 408.778], Standard Error of Mean 328.227 — Mean Difference (Final Values) = Least Squares Mean Difference

6. Secondary Outcome: Analgesics Used Post Discharge (Ibuprofen) for the Pregabalin 150 mg and Placebo Treatment Groups
Description: as for outcome 5
Time Frame: Week 2, Week 4, Week 6/ET
Population: MITT. There were not enough subjects with data at Week 2 and Week 4 for Ibuprofen to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Pregabalin (150 mg) | Placebo
Number analyzed (Participants) | 3 | 1
mg | 862.350 (584.827) | 983.850 (1119.858)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Test type: Superiority or Other; p = 0.9341, ANOVA; Mean Difference (Final Values) = -121.500, 95% CI 2-sided [-14983.36 to 14740.362], Standard Error of Mean 1169.654 — Mean Difference (Final Values) = Least Squares Mean Difference

7. Secondary Outcome: Analgesics Used Post Discharge (Ibuprofen) for the Pregabalin 300 mg Treatment Group
Description: as for outcome 5
Time Frame: Week 2, Week 4, Week 6/ET
Population: MITT. There were not enough subjects with data at Week 2 for Ibuprofen to calculate least squares mean values.
Arm/Group | Pregabalin (300 mg)
Number analyzed (Participants) | 0

8. Secondary Outcome: Analgesics Used Post Discharge (Acetylsalicylic Acid) for the Pregabalin 150 mg and Placebo Treatment Groups at Week 4
Description: Week 4 total daily dose was calculated by adding the cumulative doses during the 2 week period prior to the visit and dividing them by the number of days in the period.
Time Frame: Week 4
Population: MITT
Measure: Median (Full Range); unit: mg
Arm/Group | Pregabalin (150 mg) | Placebo
Number analyzed (Participants) | 5 | 1
mg | 650.000 (0.000) [81.000 to 1300.00] | 22.100 [22.100 to 22.100]
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 302.900, 95% CI 2-sided [302.900 to 302.900], Standard Error of Mean 0.000 — Mean Difference (Final Values) = Least Squares Mean Difference

9. Secondary Outcome: Analgesics Used Post Discharge (Acetylsalicylic Acid) for the Pregabalin 300 mg Treatment Group at Week 4
Description: as for outcome 8
Time Frame: Week 4
Arm/Group | Pregabalin (300 mg)
Number analyzed (Participants) | 0

10. Secondary Outcome: Analgesics Used Post Discharge (Acetylsalicylic Acid) for the Pregabalin 150 mg and Placebo Treatment Groups at Week 6/ET
Description: Week 6 total daily dose was calculated by adding the cumulative doses during the 2 week period prior to the visit and dividing them by the number of days in the period.
Time Frame: Week 6/ET
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Pregabalin (150 mg)
Number analyzed (Participants) | 5
mg | 513.163 (200.647)

11. Secondary Outcome: Analgesics Used Post Discharge (Acetylsalicylic Acid) for the Pregabalin 300 mg and Placebo Treatment Groups at Week 6/ET
Description: as for outcome 10
Time Frame: Week 6/ET
Population: MITT
Arm/Group | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: The Effect of Pregabalin Compared to Placebo on the Occurrence of Opioid-Related Symptoms as Assessed Using the Opioid-Related Symptom Distress Scale (OR-SDS) - Frequency Composite Score
Description: The OR-SDS was used to assess subject-reported levels of frequency concerning 10 symptoms known to be associated with opioid medication usage: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty with urination, confusion, and retching/vomiting. Symptom frequency was rated as: 1=rarely, 2=occasionally, 3=frequently, or 4=almost constantly. The average score for each symptom was calculated by taking the mean of patient-reported score. Total possible frequency score: 0 (less frequent) to 4 (more frequent).
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, Discharge, Week 2, Week 4, Week 6/ET
Population: MITT.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 87 | 86 | 81
scores on a scale
  24 hours (n=72, 69, 69) | 0.767 (0.069) | 0.808 (0.072) | 0.888 (0.074)
  48 hours (n=83, 86, 76) | 0.782 (0.061) | 0.779 (0.060) | 0.908 (0.063)
  72 hours (n=81, 77, 73) | 0.669 (0.064) | 0.688 (0.066) | 0.726 (0.069)
  96 hours (n=49, 53, 54) | 0.623 (0.087) | 0.656 (0.083) | 0.676 (0.082)
  120 hours (n=19, 17, 23) | 0.427 (0.086) | 0.405 (0.087) | 0.446 (0.087)
  Discharge (n=86, 85, 81) | 0.567 (0.056) | 0.619 (0.056) | 0.664 (0.058)
  Week 2 (n=87, 78, 79) | 0.535 (0.056) | 0.525 (0.058) | 0.513 (0.059)
  Week 4 (n=77, 69, 67) | 0.402 (0.048) | 0.415 (0.050) | 0.391 (0.053)
  Week 6/ET (n=78, 66, 71) | 0.249 (0.043) | 0.386 (0.047) | 0.239 (0.047)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.1661, ANOVA; Mean Difference (Final Values) = -0.121, 95% CI [-0.293 to 0.051], Standard Error of Mean 0.087 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.3604, ANOVA; Mean Difference (Final Values) = -0.081, 95% CI [-0.254 to 0.093], Standard Error of Mean 0.088 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.1299, ANOVA; Mean Difference (Final Values) = -0.126, 95% CI [-0.290 to 0.037], Standard Error of Mean 0.083 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.1167, ANOVA; Mean Difference (Final Values) = -0.129, 95% CI [-0.290 to 0.032], Standard Error of Mean 0.082 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.5271, ANOVA; Mean Difference (Final Values) = -0.057, 95% CI [-0.234 to 0.120], Standard Error of Mean 0.090 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.6731, ANOVA; Mean Difference (Final Values) = -0.038, 95% CI [-0.215 to 0.139], Standard Error of Mean 0.090 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.5936, ANOVA; Mean Difference (Final Values) = -0.053, 95% CI [-0.247 to 0.142], Standard Error of Mean 0.098 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.8368, ANOVA; Mean Difference (Final Values) = -0.019, 95% CI [-0.206 to 0.167], Standard Error of Mean 0.094 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.8659, ANOVA; Mean Difference (Final Values) = -0.019, 95% CI [-0.242 to 0.204], Standard Error of Mean 0.111 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.7151, ANOVA; Mean Difference (Final Values) = -0.041, 95% CI [-0.266 to 0.184], Standard Error of Mean 0.112 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.2121, ANOVA; Mean Difference (Final Values) = -0.097, 95% CI [-0.249 to 0.056], Standard Error of Mean 0.077 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5607, ANOVA; Mean Difference (Final Values) = -0.045, 95% CI [-0.197 to 0.107], Standard Error of Mean 0.077 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7797, ANOVA; Mean Difference (Final Values) = 0.022, 95% CI [-0.130 to 0.173], Standard Error of Mean 0.077 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8761, ANOVA; Mean Difference (Final Values) = 0.012, 95% CI [-0.143 to 0.167], Standard Error of Mean 0.079 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8619, ANOVA; Mean Difference (Final Values) = 0.012, 95% CI [-0.121 to 0.144], Standard Error of Mean 0.067 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.7256, ANOVA; Mean Difference (Final Values) = 0.024, 95% CI [-0.111 to 0.159], Standard Error of Mean 0.068 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8659, ANOVA; Mean Difference (Final Values) = 0.010, 95% CI [-0.110 to 0.131], Standard Error of Mean 0.061 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.0203, ANOVA; Mean Difference (Final Values) = 0.146, 95% CI [0.023 to 0.270], Standard Error of Mean 0.063 — Mean difference (final values) = Least squares mean difference

13. Secondary Outcome: The Effect of Pregabalin Compared to Placebo on the Occurrence of Opioid-Related Symptoms as Assessed Using the OR-SDS - Severity Composite Score
Description: The OR-SDS was used to assess subject-reported levels of severity concerning 10 symptoms known to be associated with opioid medication usage: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty with urination, confusion, and retching/vomiting. Symptom severity was rated as: 1=slight, 2=moderate, 3=severe, or 4=very severe. The average score for each symptom was calculated by taking the mean of patient-reported score. Total possible severity score: 0 (less severe) to 4 (more severe).
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, Discharge, Week 2, Week 4, Week 6/ET
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 87 | 86 | 82
scores on a scale
  24 hours (n=72, 69, 69) | 0.579 (0.059) | 0.590 (0.061) | 0.621 (0.062)
  48 hours (n=83, 86, 77) | 0.642 (0.051) | 0.624 (0.050) | 0.695 (0.053)
  72 hours (n=81, 77, 73) | 0.539 (0.054) | 0.534 (0.055) | 0.562 (0.057)
  96 hours (n=49, 53, 54) | 0.509 (0.070) | 0.502 (0.067) | 0.535 (0.066)
  120 hours (n=19, 17, 23) | 0.366 (0.066) | 0.334 (0.067) | 0.391 (0.066)
  Discharge (n=86, 85, 82) | 0.451 (0.048) | 0.495 (0.048) | 0.488 (0.049)
  Week 2 (n=87, 78, 79) | 0.390 (0.043) | 0.375 (0.045) | 0.364 (0.045)
  Week 4 (n=77, 69, 67) | 0.269 (0.034) | 0.308 (0.036) | 0.247 (0.037)
  Week 6/ET (n=78, 66, 71) | 0.182 (0.034) | 0.282 (0.037) | 0.175 (0.037)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.5791, ANOVA; Mean Difference (Final Values) = -0.041, 95% CI [-0.187 to 0.105], Standard Error of Mean 0.074 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.6829, ANOVA; Mean Difference (Final Values) = -0.031, 95% CI [-0.178 to 0.117], Standard Error of Mean 0.075 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.4516, ANOVA; Mean Difference (Final Values) = -0.053, 95% CI [-0.190 to 0.085], Standard Error of Mean 0.070 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.3014, ANOVA; Mean Difference (Final Values) = -0.071, 95% CI [-0.207 to 0.064], Standard Error of Mean 0.069 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.7628, ANOVA; Mean Difference (Final Values) = -0.023, 95% CI [-0.171 to 0.125], Standard Error of Mean 0.075 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.7110, ANOVA; Mean Difference (Final Values) = -0.028, 95% CI [-0.176 to 0.120], Standard Error of Mean 0.075 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.7382, ANOVA; Mean Difference (Final Values) = -0.026, 95% CI [-0.183 to 0.130], Standard Error of Mean 0.079 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.6586, ANOVA; Mean Difference (Final Values) = -0.034, 95% CI [-0.183 to 0.116], Standard Error of Mean 0.076 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.7691, ANOVA; Mean Difference (Final Values) = -0.025, 95% CI [-0.195 to 0.145], Standard Error of Mean 0.084 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.5070, ANOVA; Mean Difference (Final Values) = -0.057, 95% CI [-0.229 to 0.115], Standard Error of Mean 0.085 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5802, ANOVA; Mean Difference (Final Values) = -0.036, 95% CI [-0.166 to 0.093], Standard Error of Mean 0.066 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.9190, ANOVA; Mean Difference (Final Values) = 0.007, 95% CI [-0.122 to 0.136], Standard Error of Mean 0.065 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.6559, ANOVA; Mean Difference (Final Values) = 0.026, 95% CI [-0.090 to 0.143], Standard Error of Mean 0.059 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8552, ANOVA; Mean Difference (Final Values) = 0.011, 95% CI [-0.108 to 0.130], Standard Error of Mean 0.060 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6364, ANOVA; Mean Difference (Final Values) = 0.023, 95% CI [-0.072 to 0.117], Standard Error of Mean 0.048 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2127, ANOVA; Mean Difference (Final Values) = 0.061, 95% CI [-0.035 to 0.157], Standard Error of Mean 0.049 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8746, ANOVA; Mean Difference (Final Values) = 0.007, 95% CI [-0.086 to 0.101], Standard Error of Mean 0.047 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.0286, ANOVA; Mean Difference (Final Values) = 0.107, 95% CI [0.011 to 0.202], Standard Error of Mean 0.048 — Mean difference (final values) = Least squares mean difference

14. Secondary Outcome: The Effect of Pregabalin Compared to Placebo on the Occurrence of Opioid-Related Symptoms as Assessed Using the OR-SDS - Degree of Bother Composite Score
Description: The OR-SDS was used to assess subject-reported level of degree of bother concerning 10 symptoms known to be associated with opioid medication usage: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty with urination, confusion, and retching/vomiting. Symptom degree of bother was rated as: 1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit, or 5=very much. Average score for each symptom was calculated by taking the mean of patient-reported score. Total possible degree of bother score: 0 (less degree of bother) to 5 (greater degree of bother).
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, Discharge, Week 2, Week 4, Week 6/ET
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 87 | 86 | 82
scores on a scale
  24 hours (n=72, 69, 69) | 0.671 (0.081) | 0.788 (0.084) | 0.836 (0.086)
  48 hours (n=83, 86, 77) | 0.810 (0.067) | 0.769 (0.066) | 0.918 (0.070)
  72 hours (n=81, 77, 73) | 0.686 (0.077) | 0.694 (0.080) | 0.822 (0.083)
  96 hours (n=49, 53, 54) | 0.572 (0.096) | 0.623 (0.092) | 0.703 (0.090)
  120 hours (n=19, 17, 23) | 0.565 (0.111) | 0.439 (0.113) | 0.574 (0.113)
  Discharge (n=86, 85, 82) | 0.575 (0.067) | 0.616 (0.067) | 0.697 (0.069)
  Week 2 (n=87, 78, 79) | 0.527 (0.063) | 0.506 (0.066) | 0.533 (0.067)
  Week 4 (n=77, 69, 67) | 0.395 (0.053) | 0.433 (0.055) | 0.354 (0.058)
  Week 6/ET (n=78, 66, 71) | 0.260 (0.049) | 0.401 (0.053) | 0.274 (0.053)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.1078, ANOVA; Mean Difference (Final Values) = -0.165, 95% CI [-0.367 to 0.036], Standard Error of Mean 0.102 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.6406, ANOVA; Mean Difference (Final Values) = -0.048, 95% CI [-0.252 to 0.155], Standard Error of Mean 0.103 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.2404, ANOVA; Mean Difference (Final Values) = -0.108, 95% CI [-0.289 to 0.073], Standard Error of Mean 0.092 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.1005, ANOVA; Mean Difference (Final Values) = -0.149, 95% CI [-0.327 to 0.029], Standard Error of Mean 0.090 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.2109, ANOVA; Mean Difference (Final Values) = -0.136, 95% CI [-0.349 to 0.078], Standard Error of Mean 0.108 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.2399, ANOVA; Mean Difference (Final Values) = -0.128, 95% CI [-0.342 to 0.086], Standard Error of Mean 0.108 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.2272, ANOVA; Mean Difference (Final Values) = -0.131, 95% CI [-0.346 to 0.083], Standard Error of Mean 0.108 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.4417, ANOVA; Mean Difference (Final Values) = -0.080, 95% CI [-0.285 to 0.125], Standard Error of Mean 0.104 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.9502, ANOVA; Mean Difference (Final Values) = -0.009, 95% CI [-0.299 to 0.281], Standard Error of Mean 0.144 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.3550, ANOVA; Mean Difference (Final Values) = -0.135, 95% CI [-0.426 to 0.156], Standard Error of Mean 0.144 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1888, ANOVA; Mean Difference (Final Values) = -0.122, 95% CI [-0.304 to 0.060], Standard Error of Mean 0.092 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.3774, ANOVA; Mean Difference (Final Values) = -0.081, 95% CI [-0.262 to 0.100], Standard Error of Mean 0.092 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.9452, ANOVA; Mean Difference (Final Values) = -0.006, 95% CI [-0.178 to 0.166], Standard Error of Mean 0.087 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7663, ANOVA; Mean Difference (Final Values) = -0.026, 95% CI [-0.201 to 0.148], Standard Error of Mean 0.089 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.5777, ANOVA; Mean Difference (Final Values) = 0.041, 95% CI [-0.104 to 0.186], Standard Error of Mean 0.074 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2916, ANOVA; Mean Difference (Final Values) = 0.079, 95% CI [-0.069 to 0.227], Standard Error of Mean 0.075 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8389, ANOVA; Mean Difference (Final Values) = -0.014, 95% CI [-0.150 to 0.122], Standard Error of Mean 0.069 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.0734, ANOVA; Mean Difference (Final Values) = 0.127, 95% CI [-0.012 to 0.266], Standard Error of Mean 0.070 — Mean difference (final values) = Least squares mean difference

15. Secondary Outcome: The Effect of Pregabalin Compared to Placebo on the Occurrence of Opioid-Related Symptoms as Assessed Using the OR-SDS - Overall Composite Score
Description: The OR-SDS assessed subject-reported levels of frequency, severity and degree of bother for 10 symptoms known to be associated with opioid medication usage: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty with urination, confusion, retching and vomiting. The overall composite score was the average across frequency, severity, and degree of bother scores. Total possible score: 0 (better) to 4.34 (worse).
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, Discharge, Week 2, Week 4, Week 6/ET
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 87 | 86 | 82
scores on a scale
  24 hours (n=72, 69, 69) | 0.669 (0.067) | 0.727 (0.069) | 0.778 (0.071)
  48 hours (n=83, 86, 77) | 0.743 (0.056) | 0.722 (0.055) | 0.838 (0.059)
  72 hours (n=81, 77, 73) | 0.630 (0.063) | 0.637 (0.065) | 0.703 (0.067)
  96 hours (n=49, 53, 54) | 0.567 (0.082) | 0.593 (0.079) | 0.637 (0.077)
  120 hours (n=19, 17, 23) | 0.453 (0.084) | 0.393 (0.086) | 0.471 (0.085)
  Discharge (n=86, 85, 82) | 0.530 (0.055) | 0.575 (0.055) | 0.615 (0.056)
  Week 2 (n=87, 78, 79) | 0.482 (0.052) | 0.467 (0.055) | 0.469 (0.056)
  Week 4 (n=77, 69, 67) | 0.354 (0.044) | 0.384 (0.046) | 0.329 (0.048)
  Week 6/ET (n=78, 66, 71) | 0.230 (0.041) | 0.355 (0.045) | 0.229 (0.045)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.1949, ANOVA; Mean Difference (Final Values) = -0.110, 95% CI [-0.276 to 0.057], Standard Error of Mean 0.084 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.5431, ANOVA; Mean Difference (Final Values) = -0.052, 95% CI [-0.220 to 0.116], Standard Error of Mean 0.085 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.2164, ANOVA; Mean Difference (Final Values) = -0.095, 95% CI [-0.247 to 0.056], Standard Error of Mean 0.077 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.1251, ANOVA; Mean Difference (Final Values) = -0.117, 95% CI [-0.266 to 0.033], Standard Error of Mean 0.076 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.4079, ANOVA; Mean Difference (Final Values) = -0.073, 95% CI [-0.247 to 0.101], Standard Error of Mean 0.088 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.4562, ANOVA; Mean Difference (Final Values) = -0.066, 95% CI [-0.240 to 0.108], Standard Error of Mean 0.088 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.4526, ANOVA; Mean Difference (Final Values) = -0.070, 95% CI [-0.254 to 0.114], Standard Error of Mean 0.093 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.6186, ANOVA; Mean Difference (Final Values) = -0.045, 95% CI [-0.221 to 0.132], Standard Error of Mean 0.089 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.8712, ANOVA; Mean Difference (Final Values) = -0.018, 95% CI [-0.237 to 0.202], Standard Error of Mean 0.109 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.4784, ANOVA; Mean Difference (Final Values) = -0.078, 95% CI [-0.300 to 0.143], Standard Error of Mean 0.110 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.2635, ANOVA; Mean Difference (Final Values) = -0.084, 95% CI [-0.232 to 0.064], Standard Error of Mean 0.075 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.6009, ANOVA; Mean Difference (Final Values) = -0.039, 95% CI [-0.187 to 0.108], Standard Error of Mean 0.075 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8559, ANOVA; Mean Difference (Final Values) = 0.013, 95% CI [-0.130 to 0.156], Standard Error of Mean 0.073 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.9841, ANOVA; Mean Difference (Final Values) = -0.001, 95% CI [-0.147 to 0.144], Standard Error of Mean 0.074 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6771, ANOVA; Mean Difference (Final Values) = 0.025, 95% CI [-0.095 to 0.146], Standard Error of Mean 0.061 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.3717, ANOVA; Mean Difference (Final Values) = 0.056, 95% CI [-0.067 to 0.178], Standard Error of Mean 0.062 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9863, ANOVA; Mean Difference (Final Values) = 0.001, 95% CI [-0.114 to 0.116], Standard Error of Mean 0.058 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.0355, ANOVA; Mean Difference (Final Values) = 0.126, 95% CI [0.009 to 0.243], Standard Error of Mean 0.059 — Mean difference (final values) = Least squares mean difference

16. Secondary Outcome: Total Clinically Meaningful Event (CME) Score
Description: CMEs were defined using OR-SDS (assesses subject-reported levels of severity concerning 10 symptoms associated with opioid medication usage: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty with urination, confusion and retching/vomiting). CME = any symptom rated as severe or very severe, with the exception of confusion. Confusion was defined as a CME if the severity score was at least moderate. Total score = the sum of CMEs across symptoms. Each CME = 1 point. Total CME score ranges from 0 to 9.
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, Discharge, Week 2, Week 4, and Week 6/ET
Population: MITT.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 87 | 86 | 82
scores on a scale
  24 hours (n=72, 69, 69) | 0.822 (0.161) | 0.817 (0.166) | 0.772 (0.171)
  48 hours (n=83, 86, 87) | 0.814 (0.141) | 0.834 (0.138) | 0.789 (0.146)
  72 hours (n=81, 77, 73) | 0.647 (0.134) | 0.570 (0.138) | 0.613 (0.144)
  96 hours (n=49, 53, 54) | 0.440 (0.173) | 0.489 (0.164) | 0.284 (0.162)
  120 hours (n=19, 17, 23) | 0.178 (0.089) | 0.350 (0.091) | 0.246 (0.090)
  Discharge (n=86, 85, 82) | 0.429 (0.113) | 0.502 (0.114) | 0.352 (0.117)
  Week 2 (n=87, 78, 79) | 0.328 (0.093) | 0.311 (0.097) | 0.171 (0.099)
  Week 4 (n=77, 69, 67) | 0.116 (0.059) | 0.236 (0.062) | 0.032 (0.064)
  Week 6/ET (n=78, 66, 71) | 0.059 (0.062) | 0.260 (0.068) | 0.051 (0.067)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.8071, ANOVA; Mean Difference (Final Values) = 0.049, 95% CI [-0.350 to 0.449], Standard Error of Mean 0.202 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.8282, ANOVA; Mean Difference (Final Values) = 0.044, 95% CI [-0.359 to 0.447], Standard Error of Mean 0.204 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.8972, ANOVA; Mean Difference (Final Values) = 0.025, 95% CI [-0.353 to 0.403], Standard Error of Mean 0.192 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.8159, ANOVA; Mean Difference (Final Values) = 0.044, 95% CI [-0.329 to 0.418], Standard Error of Mean 0.190 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.8577, ANOVA; Mean Difference (Final Values) = 0.034, 95% CI [-0.337 to 0.405], Standard Error of Mean 0.188 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.8158, ANOVA; Mean Difference (Final Values) = -0.044, 95% CI [-0.415 to 0.327], Standard Error of Mean 0.188 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.4243, ANOVA; Mean Difference (Final Values) = 0.156, 95% CI [-0.229 to 0.541], Standard Error of Mean 0.195 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.2742, ANOVA; Mean Difference (Final Values) = 0.205, 95% CI [-0.164 to 0.574], Standard Error of Mean 0.187 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.5569, ANOVA; Mean Difference (Final Values) = -0.069, 95% CI [-0.302 to 0.165], Standard Error of Mean 0.116 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.3762, ANOVA; Mean Difference (Final Values) = 0.103, 95% CI [-0.130 to 0.336], Standard Error of Mean 0.116 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.6203, ANOVA; Mean Difference (Final Values) = 0.077, 95% CI [-0.229 to 0.383], Standard Error of Mean 0.155 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.3343, ANOVA; Mean Difference (Final Values) = 0.150, 95% CI [-0.155 to 0.455], Standard Error of Mean 0.155 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2213, ANOVA; Mean Difference (Final Values) = 0.157, 95% CI [-0.096 to 0.410], Standard Error of Mean 0.128 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2863, ANOVA; Mean Difference (Final Values) = 0.140, 95% CI [-0.118 to 0.399], Standard Error of Mean 0.131 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.3050, ANOVA; Mean Difference (Final Values) = 0.084, 95% CI [-0.077 to 0.245], Standard Error of Mean 0.082 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0155, ANOVA; Mean Difference (Final Values) = 0.204, 95% CI [0.039 to 0.368], Standard Error of Mean 0.083 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9243, ANOVA; Mean Difference (Final Values) = 0.008, 95% CI [-0.164 to 0.181], Standard Error of Mean 0.087 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.0201, ANOVA; Mean Difference (Final Values) = 0.210, 95% CI [0.033 to 0.386], Standard Error of Mean 0.089 — Mean difference (final values) = Least squares mean difference

17. Secondary Outcome: Pain Interference Index Score as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Pain interference index = average of pain interference question (Q) 5A to 5G. Questions were asked as follows: how, during the past 24 hours, has pain interfered with general activity (Q5A), mood (Q5B), walking ability (Q5C), normal work (outside home and housework) (Q5D), relations with other people (Q5E), sleep (Q5F), enjoyment of life (Q5G). Scale: 0=does not interfere to 10=completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 80 | 80
scores on a scale
  Discharge (n=83, 80, 74) | 3.427 (0.230) | 3.488 (0.230) | 3.887 (0.246)
  Week 2 (n=86, 78, 80) | 2.969 (0.236) | 2.814 (0.245) | 3.037 (0.251)
  Week 4 (n=77, 69, 67) | 2.162 (0.202) | 1.996 (0.208) | 2.094 (0.224)
  Week 6/ET (n=78, 67, 71) | 1.597 (0.199) | 1.637 (0.214) | 1.662 (0.215)
  Month 3 (n=30, 32, 35) | 1.139 (0.367) | 1.335 (0.375) | 1.629 (0.366)
  Month 6 (n=31, 25, 27) | 1.513 (0.264) | 1.300 (0.241) | 0.852 (0.253)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1537, ANOVA; Mean Difference (Final Values) = -0.460, 95% CI [-1.093 to 0.173], Standard Error of Mean 0.321 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.2208, ANOVA; Mean Difference (Final Values) = -0.398, 95% CI [-1.038 to 0.241], Standard Error of Mean 0.324 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8355, ANOVA; Mean Difference (Final Values) = -0.068, 95% CI [-0.707 to 0.572], Standard Error of Mean 0.325 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.5024, ANOVA; Mean Difference (Final Values) = -0.222, 95% CI [-0.875 to 0.430], Standard Error of Mean 0.331 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8116, ANOVA; Mean Difference (Final Values) = 0.067, 95% CI [-0.489 to 0.624], Standard Error of Mean 0.282 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.7325, ANOVA; Mean Difference (Final Values) = -0.099, 95% CI [-0.667 to 0.469], Standard Error of Mean 0.288 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8133, ANOVA; Mean Difference (Final Values) = -0.066, 95% CI [-0.614 to 0.482], Standard Error of Mean 0.278 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9307, ANOVA; Mean Difference (Final Values) = -0.025, 95% CI [-0.588 to 0.538], Standard Error of Mean 0.285 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.2682, ANOVA; Mean Difference (Final Values) = -0.490, 95% CI [-1.364 to 0.385], Standard Error of Mean 0.439 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.4784, ANOVA; Mean Difference (Final Values) = -0.294, 95% CI [-1.116 to 0.528], Standard Error of Mean 0.413 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.0255, ANOVA; Mean Difference (Final Values) = 0.661, 95% CI [0.084 to 1.239], Standard Error of Mean 0.298 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.1591, ANOVA; Mean Difference (Final Values) = 0.448, 95% CI [-0.180 to 1.076], Standard Error of Mean 0.314 — Mean difference (final values) = Least squares mean difference

18. Secondary Outcome: Pain Interference With Relations With People as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Q5E: Subject response to 'how, during the past 24 hours, pain has interfered with your relations with other people'. Scale: 0 = does not interfere to 10 = completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 80 | 80
scores on a scale
  Discharge (n=83, 80, 74) | 1.837 (0.266) | 1.716 (0.266) | 2.624 (0.284)
  Week 2 (n=86, 78, 80) | 1.566 (0.231) | 1.370 (0.240) | 1.671 (0.246)
  Week 4 (n=77, 69, 67) | 1.004 (0.215) | 1.162 (0.222) | 1.187 (0.238)
  Week 6/ET (n=78, 67, 71) | 0.544 (0.171) | 0.845 (0.184) | 0.898 (0.185)
  Month 3 (n=30, 32, 35) | 0.253 (0.377) | 0.861 (0.377) | 1.364 (0.365)
  Month 6 (n=31, 25, 27) | 0.802 (0.245) | 1.060 (0.226) | 0.626 (0.235)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0359, ANOVA; Mean Difference (Final Values) = -0.786, 95% CI [-1.520 to -0.052], Standard Error of Mean 0.372 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0161, ANOVA; Mean Difference (Final Values) = -0.907, 95% CI [-1.644 to -0.170], Standard Error of Mean 0.374 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7416, ANOVA; Mean Difference (Final Values) = -0.105, 95% CI [-0.733 to 0.523], Standard Error of Mean 0.319 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.3527, ANOVA; Mean Difference (Final Values) = -0.301, 95% CI [-0.939 to 0.336], Standard Error of Mean 0.324 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.5419, ANOVA; Mean Difference (Final Values) = -0.184, 95% CI [-0.776 to 0.409], Standard Error of Mean 0.300 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9333, ANOVA; Mean Difference (Final Values) = -0.026, 95% CI [-0.628 to 0.577], Standard Error of Mean 0.305 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.1420, ANOVA; Mean Difference (Final Values) = -0.354, 95% CI [-0.827 to 0.120], Standard Error of Mean 0.240 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8290, ANOVA; Mean Difference (Final Values) = -0.053, 95% CI [-0.535 to 0.429], Standard Error of Mean 0.245 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.0138, ANOVA; Mean Difference (Final Values) = -1.111, 95% CI [-1.989 to -0.233], Standard Error of Mean 0.441 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.2300, ANOVA; Mean Difference (Final Values) = -0.503, 95% CI [-1.332 to 0.325], Standard Error of Mean 0.416 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.5151, ANOVA; Mean Difference (Final Values) = 0.175, 95% CI [-0.360 to 0.711], Standard Error of Mean 0.268 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.1460, ANOVA; Mean Difference (Final Values) = 0.433, 95% CI [-0.155 to 1.022], Standard Error of Mean 0.295 — Mean difference (final values) = Least squares mean difference

19. Secondary Outcome: Pain Interference With Enjoyment of Life as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Q5G: Subject response to 'how, during the past 24 hours, pain has interfered with your enjoyment of life'. Scale: 0 = does not interfere to 10 = completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 80 | 80
scores on a scale
  Discharge (n=83, 80, 74) | 3.487 (0.330) | 3.769 (0.330) | 3.744 (0.354)
  Week 2 (n=86, 78, 80) | 2.945 (0.313) | 2.802 (0.325) | 2.953 (0.334)
  Week 4 (n=77, 69, 67) | 2.152 (0.260) | 2.042 (0.268) | 1.768 (0.289)
  Week 6/ET (n=78, 67, 71) | 1.535 (0.247) | 1.720 (0.266) | 1.696 (0.267)
  Month 3 (n=30, 32, 35) | 0.944 (0.497) | 1.467 (0.513) | 1.368 (0.509)
  Month 6 (n=31, 25, 27) | 1.657 (0.404) | 1.658 (0.367) | 0.663 (0.389)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5786, ANOVA; Mean Difference (Final Values) = -0.258, 95% CI [-1.170 to 0.655], Standard Error of Mean 0.463 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.9570, ANOVA; Mean Difference (Final Values) = 0.025, 95% CI [-0.895 to 0.946], Standard Error of Mean 0.467 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.9860, ANOVA; Mean Difference (Final Values) = -0.008, 95% CI [-0.862 to 0.847], Standard Error of Mean 0.434 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7336, ANOVA; Mean Difference (Final Values) = -0.151, 95% CI [-1.021 to 0.720], Standard Error of Mean 0.442 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2939, ANOVA; Mean Difference (Final Values) = 0.384, 95% CI [-0.336 to 1.104], Standard Error of Mean 0.365 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.4615, ANOVA; Mean Difference (Final Values) = 0.274, 95% CI [-0.459 to 1.008], Standard Error of Mean 0.372 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.6433, ANOVA; Mean Difference (Final Values) = -0.161, 95% CI [-0.845 to 0.523], Standard Error of Mean 0.347 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9466, ANOVA; Mean Difference (Final Values) = 0.024, 95% CI [-0.678 to 0.726], Standard Error of Mean 0.356 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.4967, ANOVA; Mean Difference (Final Values) = -0.424, 95% CI [-1.660 to 0.812], Standard Error of Mean 0.621 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.8659, ANOVA; Mean Difference (Final Values) = 0.099, 95% CI [-1.060 to 1.257], Standard Error of Mean 0.582 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.0311, ANOVA; Mean Difference (Final Values) = 0.994, 95% CI [0.093 to 1.895], Standard Error of Mean 0.451 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.0441, ANOVA; Mean Difference (Final Values) = 0.995, 95% CI [0.027 to 1.962], Standard Error of Mean 0.485 — Mean difference (final values) = Least squares mean difference

20. Secondary Outcome: Pain Interference With General Activity as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Q5A: Subject response to 'how, during the past 24 hours, pain has interfered with your general activity. Scale: 0 = does not interfere to 10 = completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 80 | 80
scores on a scale
  Discharge (n=83, 80, 74) | 3.794 (0.317) | 4.499 (0.315) | 4.764 (0.336)
  Week 2 (n=86, 78, 80) | 3.254 (0.278) | 3.526 (0.288) | 3.524 (0.294)
  Week 4 (n=77, 69, 67) | 2.470 (0.237) | 2.417 (0.244) | 2.427 (0.260)
  Week 6/ET (n=78, 67, 71) | 2.109 (0.245) | 1.902 (0.263) | 2.028 (0.263)
  Month 3 (n=30, 32, 35) | 1.861 (0.505) | 1.547 (0.507) | 1.969 (0.492)
  Month 6 (n=31, 25, 27) | 1.738 (0.412) | 1.717 (0.376) | 1.410 (0.394)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0284, ANOVA; Mean Difference (Final Values) = -0.969, 95% CI [-1.835 to -0.104], Standard Error of Mean 0.439 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5516, ANOVA; Mean Difference (Final Values) = -0.265, 95% CI [-1.141 to 0.611], Standard Error of Mean 0.444 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4790, ANOVA; Mean Difference (Final Values) = -0.270, 95% CI [-1.020 to 0.480], Standard Error of Mean 0.380 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.9947, ANOVA; Mean Difference (Final Values) = 0.003, 95% CI [-0.765 to 0.770], Standard Error of Mean 0.390 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8943, ANOVA; Mean Difference (Final Values) = 0.044, 95% CI [-0.605 to 0.692], Standard Error of Mean 0.329 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9767, ANOVA; Mean Difference (Final Values) = -0.010, 95% CI [-0.674 to 0.654], Standard Error of Mean 0.336 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8117, ANOVA; Mean Difference (Final Values) = 0.081, 95% CI [-0.590 to 0.752], Standard Error of Mean 0.340 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.7216, ANOVA; Mean Difference (Final Values) = -0.125, 95% CI [-0.818 to 0.567], Standard Error of Mean 0.351 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.8558, ANOVA; Mean Difference (Final Values) = -0.108, 95% CI [-1.286 to 1.070], Standard Error of Mean 0.592 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.4501, ANOVA; Mean Difference (Final Values) = -0.422, 95% CI [-1.530 to 0.685], Standard Error of Mean 0.556 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.4682, ANOVA; Mean Difference (Final Values) = 0.328, 95% CI [-0.570 to 1.227], Standard Error of Mean 0.450 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.5347, ANOVA; Mean Difference (Final Values) = 0.307, 95% CI [-0.675 to 1.289], Standard Error of Mean 0.492 — Mean difference (final values) = Least squares mean difference

21. Secondary Outcome: Pain Interference With Mood as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Q5B: Subject response to 'how, during the past 24 hours, pain has interfered with your mood'. Scale: 0 = does not interfere to 10 = completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 80 | 80
scores on a scale
  Discharge (n=83, 80, 74) | 2.588 (0.292) | 2.418 (0.291) | 3.354 (0.310)
  Week 2 (n=86, 78, 80) | 2.640 (0.292) | 2.115 (0.303) | 2.554 (0.308)
  Week 4 (n=77, 69, 67) | 1.590 (0.253) | 1.511 (0.261) | 1.530 (0.279)
  Week 6/ET (n=78, 67, 71) | 1.053 (0.230) | 1.171 (0.247) | 1.325 (0.247)
  Month 3 (n=30, 32, 35) | 0.632 (0.328) | 0.956 (0.339) | 1.334 (0.322)
  Month 6 (n=31, 25, 27) | 1.201 (0.326) | 0.832 (0.297) | 0.369 (0.313)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0613, ANOVA; Mean Difference (Final Values) = -0.765, 95% CI [-1.568 to 0.037], Standard Error of Mean 0.407 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0230, ANOVA; Mean Difference (Final Values) = -0.936, 95% CI [-1.741 to -0.130], Standard Error of Mean 0.409 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8306, ANOVA; Mean Difference (Final Values) = 0.086, 95% CI [-0.703 to 0.875], Standard Error of Mean 0.400 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2814, ANOVA; Mean Difference (Final Values) = -0.439, 95% CI [-1.242 to 0.363], Standard Error of Mean 0.407 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8637, ANOVA; Mean Difference (Final Values) = 0.061, 95% CI [-0.636 to 0.757], Standard Error of Mean 0.353 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9585, ANOVA; Mean Difference (Final Values) = -0.019, 95% CI [-0.727 to 0.689], Standard Error of Mean 0.359 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.3975, ANOVA; Mean Difference (Final Values) = -0.272, 95% CI [-0.906 to 0.361], Standard Error of Mean 0.321 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.6386, ANOVA; Mean Difference (Final Values) = -0.154, 95% CI [-0.799 to 0.491], Standard Error of Mean 0.327 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.0813, ANOVA; Mean Difference (Final Values) = -0.702, 95% CI [-1.493 to 0.089], Standard Error of Mean 0.397 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.3100, ANOVA; Mean Difference (Final Values) = -0.378, 95% CI [-1.114 to 0.358], Standard Error of Mean 0.370 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.0231, ANOVA; Mean Difference (Final Values) = 0.831, 95% CI [0.118 to 1.545], Standard Error of Mean 0.357 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.2367, ANOVA; Mean Difference (Final Values) = 0.463, 95% CI [-0.311 to 1.237], Standard Error of Mean 0.388 — Mean difference (final values) = Least squares mean difference

22. Secondary Outcome: Pain Interference With Walking Ability as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Q5C: Subject response to 'how, during the past 24 hours, pain has interfered with your walking ability'. Scale: 0 = does not interfere to 10 = completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 80 | 80
scores on a scale
  Discharge (n=83, 80, 74) | 4.918 (0.320) | 4.728 (0.319) | 4.982 (0.342)
  Week 2 (n=86, 78, 80) | 3.297 (0.278) | 3.344 (0.289) | 3.425 (0.296)
  Week 4 (n=77, 69, 67) | 2.646 (0.259) | 2.108 (0.267) | 2.442 (0.286)
  Week 6/ET (n=78, 67, 71) | 2.004 (0.237) | 1.886 (0.254) | 1.742 (0.256)
  Month 3 (n=30, 32, 35) | 1.439 (0.419) | 1.907 (0.434) | 1.928 (0.414)
  Month 6 (n=31, 25, 27) | 1.573 (0.322) | 1.391 (0.293) | 1.126 (0.308)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.8868, ANOVA; Mean Difference (Final Values) = -0.064, 95% CI [-0.947 to 0.820], Standard Error of Mean 0.448 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5733, ANOVA; Mean Difference (Final Values) = -0.254, 95% CI [-1.142 to 0.634], Standard Error of Mean 0.450 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7385, ANOVA; Mean Difference (Final Values) = -0.128, 95% CI [-0.884 to 0.628], Standard Error of Mean 0.384 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8353, ANOVA; Mean Difference (Final Values) = -0.081, 95% CI [-0.849 to 0.687], Standard Error of Mean 0.390 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.5737, ANOVA; Mean Difference (Final Values) = 0.204, 95% CI [-0.510 to 0.918], Standard Error of Mean 0.362 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.3640, ANOVA; Mean Difference (Final Values) = -0.335, 95% CI [-1.060 to 0.391], Standard Error of Mean 0.368 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.4315, ANOVA; Mean Difference (Final Values) = 0.262, 95% CI [-0.393 to 0.917], Standard Error of Mean 0.332 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.6727, ANOVA; Mean Difference (Final Values) = 0.143, 95% CI [-0.525 to 0.812], Standard Error of Mean 0.339 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.3361, ANOVA; Mean Difference (Final Values) = -0.489, 95% CI [-1.496 to 0.517], Standard Error of Mean 0.505 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.9634, ANOVA; Mean Difference (Final Values) = -0.022, 95% CI [-0.955 to 0.912], Standard Error of Mean 0.469 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.2098, ANOVA; Mean Difference (Final Values) = 0.446, 95% CI [-0.257 to 1.150], Standard Error of Mean 0.352 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.4900, ANOVA; Mean Difference (Final Values) = 0.265, 95% CI [-0.497 to 1.027], Standard Error of Mean 0.382 — Mean difference (final values) = Least squares mean difference

23. Secondary Outcome: Pain Interference With Normal Work as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Q5D: Subject response to 'how, during the past 24 hours, pain has interfered with your normal work (work outside the home and housework)'. Scale: 0 = does not interfere to 10 = completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 78 | 79
scores on a scale
  Discharge (n=82, 77, 72) | 4.879 (0.390) | 4.738 (0.395) | 4.873 (0.418)
  Week 2 (n=86, 78, 79) | 4.010 (0.335) | 3.539 (0.347) | 3.831 (0.355)
  Week 4 (n=77, 69, 67) | 2.833 (0.275) | 2.500 (0.285) | 2.895 (0.305)
  Week 6/ET (n=78, 67, 71) | 2.133 (0.269) | 2.152 (0.291) | 2.040 (0.291)
  Month 3 (n=30, 32, 35) | 1.797 (0.510) | 1.731 (0.520) | 2.264 (0.507)
  Month 6 (n=31, 25, 27) | 1.627 (0.288) | 1.349 (0.263) | 1.029 (0.276)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.9912, ANOVA; Mean Difference (Final Values) = 0.006, 95% CI [-1.070 to 1.082], Standard Error of Mean 0.546 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.8076, ANOVA; Mean Difference (Final Values) = -0.135, 95% CI [-1.227 to 0.957], Standard Error of Mean 0.554 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.6978, ANOVA; Mean Difference (Final Values) = 0.179, 95% CI [-0.727 to 1.085], Standard Error of Mean 0.460 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.5344, ANOVA; Mean Difference (Final Values) = -0.293, 95% CI [-1.219 to 0.634], Standard Error of Mean 0.470 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8721, ANOVA; Mean Difference (Final Values) = -0.062, 95% CI [-0.819 to 0.695], Standard Error of Mean 0.384 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.3179, ANOVA; Mean Difference (Final Values) = -0.395, 95% CI [-1.173 to 0.383], Standard Error of Mean 0.394 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8037, ANOVA; Mean Difference (Final Values) = 0.094, 95% CI [-0.648 to 0.835], Standard Error of Mean 0.376 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.7731, ANOVA; Mean Difference (Final Values) = 0.113, 95% CI [-0.656 to 0.881], Standard Error of Mean 0.390 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.4461, ANOVA; Mean Difference (Final Values) = -0.468, 95% CI [-1.684 to 0.748], Standard Error of Mean 0.611 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.3568, ANOVA; Mean Difference (Final Values) = -0.533, 95% CI [-1.679 to 0.612], Standard Error of Mean 0.575 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.0623, ANOVA; Mean Difference (Final Values) = 0.598, 95% CI [-0.032 to 1.227], Standard Error of Mean 0.315 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.3529, ANOVA; Mean Difference (Final Values) = 0.320, 95% CI [-0.364 to 1.005], Standard Error of Mean 0.343 — Mean difference (final values) = Least squares mean difference

24. Secondary Outcome: Pain Interference With Sleep as Measured by the m-BPI-sf
Description: m-BPI-sf questionnaire (7-items) assessed pain interference with functional activities during the past 24 hours. Q5F: Subject response to 'how, during the past 24 hours, pain has interfered with your sleep'. Scale: 0 = does not interfere to 10 = completely interferes.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET, Month 3, Month 6
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 80 | 80
scores on a scale
  Discharge (n=83, 80, 74) | 2.696 (0.299) | 2.642 (0.299) | 3.307 (0.318)
  Week 2 (n=86, 78, 80) | 3.139 (0.333) | 3.015 (0.345) | 3.587 (0.353)
  Week 4 (n=77, 69, 67) | 2.478 (0.278) | 2.166 (0.288) | 2.668 (0.308)
  Week 6/ET (n=78, 67, 71) | 1.847 (0.275) | 1.701 (0.296) | 2.070 (0.296)
  Month 3 (n=30, 32, 35) | 1.276 (0.537) | 0.941 (0.548) | 1.499 (0.526)
  Month 6 (n=31, 25, 27) | 1.963 (0.482) | 1.005 (0.439) | 0.778 (0.464)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1448, ANOVA; Mean Difference (Final Values) = -0.611, 95% CI [-1.434 to 0.212], Standard Error of Mean 0.417 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1148, ANOVA; Mean Difference (Final Values) = -0.665, 95% CI [-1.494 to 0.163], Standard Error of Mean 0.420 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.3285, ANOVA; Mean Difference (Final Values) = -0.448, 95% CI [-1.350 to 0.454], Standard Error of Mean 0.458 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2205, ANOVA; Mean Difference (Final Values) = -0.572, 95% CI [-1.490 to 0.346], Standard Error of Mean 0.466 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6266, ANOVA; Mean Difference (Final Values) = -0.190, 95% CI [-0.958 to 0.578], Standard Error of Mean 0.389 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2077, ANOVA; Mean Difference (Final Values) = -0.502, 95% CI [-1.284 to 0.281], Standard Error of Mean 0.397 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.5626, ANOVA; Mean Difference (Final Values) = -0.223, 95% CI [-0.982 to 0.536], Standard Error of Mean 0.385 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.3507, ANOVA; Mean Difference (Final Values) = -0.368, 95% CI [-1.145 to 0.408], Standard Error of Mean 0.394 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.7276, ANOVA; Mean Difference (Final Values) = -0.224, 95% CI [-1.498 to 1.050], Standard Error of Mean 0.640 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.3530, ANOVA; Mean Difference (Final Values) = -0.558, 95% CI [-1.748 to 0.631], Standard Error of Mean 0.598 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.0283, ANOVA; Mean Difference (Final Values) = 1.186, 95% CI [0.130 to 2.242], Standard Error of Mean 0.529 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.6934, ANOVA; Mean Difference (Final Values) = 0.227, 95% CI [-0.918 to 1.372], Standard Error of Mean 0.573 — Mean difference (final values) = Least squares mean difference

25. Secondary Outcome: Daily and Weekly Worst Pain During the Hospital Stay and Post Discharge Assessed by the Pain Numerical Rating Scale (NRS)
Description: Subject rated scale for worst pain over the last 24 hours. Scores ranged from 0 (no pain) to 10 (pain as bad as you can imagine). Weekly mean scores were calculated post-discharge.
Time Frame: 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours, 168 hours, and 192 hours during the hospital stay, Week 2, Week 4, Week 6/ET
Population: MITT. There were not enough subjects with data at 144, 168, and 192 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 82 | 79 | 74
scores on a scale
  12 hours (n=29, 28, 28) | 7.217 (0.597) | 7.002 (0.649) | 8.770 (0.635)
  24 hours (n=82, 79, 74) | 7.477 (0.298) | 7.290 (0.301) | 7.201 (0.311)
  48 hours (n=78, 82, 75) | 7.041 (0.267) | 6.740 (0.264) | 7.079 (0.279)
  72 hours (n=56, 52, 55) | 6.322 (0.333) | 5.977 (0.350) | 5.964 (0.343)
  96 hours (n=20, 21, 26) | 6.703 (0.624) | 4.711 (0.618) | 6.556 (0.598)
  120 hours (n=5, 3, 9) | 5.915 (0.819) | 4.346 (1.446) | 7.056 (0.663)
  Week 2 (n=79, 72, 72) | 5.255 (0.209) | 5.592 (0.223) | 5.396 (0.229)
  Week 4 (n=76, 65, 67) | 4.134 (0.220) | 4.043 (0.241) | 4.280 (0.247)
  Week 6/ET (n=61, 55, 59) | 3.455 (0.267) | 3.425 (0.276) | 3.350 (0.292)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 12 hours; Test type: Superiority or Other; p = 0.0476, ANOVA; Mean Difference (Final Values) = -1.553, 95% CI [-3.089 to -0.017], Standard Error of Mean 0.770 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 12 hours; Test type: Superiority or Other; p = 0.0237, ANOVA; Mean Difference (Final Values) = -1.768, 95% CI [-3.293 to -0.243], Standard Error of Mean 0.764 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.4925, ANOVA; Mean Difference (Final Values) = 0.276, 95% CI [-0.516 to 1.069], Standard Error of Mean 0.402 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.8299, ANOVA; Mean Difference (Final Values) = 0.089, 95% CI [-0.727 to 0.905], Standard Error of Mean 0.414 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.9185, ANOVA; Mean Difference (Final Values) = -0.038, 95% CI [-0.766 to 0.691], Standard Error of Mean 0.370 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.3619, ANOVA; Mean Difference (Final Values) = -0.339, 95% CI [-1.070 to 0.392], Standard Error of Mean 0.371 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.4309, ANOVA; Mean Difference (Final Values) = 0.358, 95% CI [-0.538 to 1.254], Standard Error of Mean 0.453 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.9778, ANOVA; Mean Difference (Final Values) = 0.013, 95% CI [-0.895 to 0.921], Standard Error of Mean 0.459 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.8503, ANOVA; Mean Difference (Final Values) = 0.147, 95% CI [-1.411 to 1.706], Standard Error of Mean 0.777 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.0183, ANOVA; Mean Difference (Final Values) = -1.845, 95% CI [-3.364 to -0.326], Standard Error of Mean 0.757 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.2860, ANOVA; Mean Difference (Final Values) = -1.141, 95% CI [-3.598 to 1.316], Standard Error of Mean 0.956 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.2040, ANOVA; Mean Difference (Final Values) = -2.710, 95% CI [-7.479 to 2.060], Standard Error of Mean 1.856 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.6332, ANOVA; Mean Difference (Final Values) = -0.141, 95% CI [-0.722 to 0.440], Standard Error of Mean 0.295 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.5183, ANOVA; Mean Difference (Final Values) = 0.196, 95% CI [-0.402 to 0.794], Standard Error of Mean 0.303 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6341, ANOVA; Mean Difference (Final Values) = -0.146, 95% CI [-0.750 to 0.458], Standard Error of Mean 0.306 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.4607, ANOVA; Mean Difference (Final Values) = -0.236, 95% CI [-0.868 to 0.395], Standard Error of Mean 0.320 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.7499, ANOVA; Mean Difference (Final Values) = 0.104, 95% CI [-0.541 to 0.750], Standard Error of Mean 0.327 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.8231, ANOVA; Mean Difference (Final Values) = 0.075, 95% CI [-0.584 to 0.733], Standard Error of Mean 0.333 — Mean difference (final values) = Least squares mean difference

26. Secondary Outcome: Daily and Weekly Average Pain During the Hospital Stay and Post Discharge Assessed by the Pain NRS
Description: Subject rated scale for average pain intensity over the last 24 hours. Scores range from 0 (no pain) to 10 (pain as bad as you can imagine). Weekly mean scores were calculated post-discharge.
Time Frame: as for outcome 25
Population: MITT. There were not enough subjects with data at 144, 168, and 192 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 85 | 84 | 82
scores on a scale
  12 hours (n=29, 28, 28) | 5.712 (0.550) | 4.845 (0.593) | 6.748 (0.600)
  24 hours (n=81, 79, 74) | 4.961 (0.255) | 4.614 (0.257) | 4.918 (0.266)
  48 hours (n=78, 82, 75) | 4.518 (0.238) | 4.309 (0.236) | 4.515 (0.249)
  72 hours (n=56, 51, 55) | 4.281 (0.280) | 3.740 (0.298) | 4.186 (0.290)
  96 hours (n=20, 21, 26) | 4.842 (0.514) | 3.126 (0.503) | 4.741 (0.488)
  120 hours (n=5, 3, 9) | 4.211 (1.002) | 2.940 (1.566) | 4.287 (0.759)
  Week 2 (n=79, 72, 71) | 3.691 (0.186) | 3.974 (0.198) | 3.987 (0.206)
  Week 4 (n=76, 65, 67) | 2.956 (0.180) | 2.845 (0.197) | 3.163 (0.203)
  Week 6/ET (n=60, 54, 59) | 2.374 (0.215) | 2.385 (0.225) | 2.389 (0.234)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 12 hours; Test type: Superiority or Other; p = 0.1486, ANOVA; Mean Difference (Final Values) = -1.036, 95% CI [-2.452 to 0.379], Standard Error of Mean 0.709 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 12 hours; Test type: Superiority or Other; p = 0.0089, ANOVA; Mean Difference (Final Values) = -1.903, 95% CI [-3.311 to -0.494], Standard Error of Mean 0.706 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.8995, ANOVA; Mean Difference (Final Values) = 0.044, 95% CI [-0.635 to 0.722], Standard Error of Mean 0.344 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.3918, ANOVA; Mean Difference (Final Values) = -0.303, 95% CI [-1.000 to 0.394], Standard Error of Mean 0.354 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.9942, ANOVA; Mean Difference (Final Values) = 0.002, 95% CI [-0.648 to 0.652], Standard Error of Mean 0.330 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.5352, ANOVA; Mean Difference (Final Values) = -0.206, 95% CI [-0.859 to 0.448], Standard Error of Mean 0.332 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.8055, ANOVA; Mean Difference (Final Values) = 0.094, 95% CI [-0.662 to 0.850], Standard Error of Mean 0.382 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.2560, ANOVA; Mean Difference (Final Values) = -0.446, 95% CI [-1.220 to 0.327], Standard Error of Mean 0.391 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.8744, ANOVA; Mean Difference (Final Values) = 0.102, 95% CI [-1.184 to 1.387], Standard Error of Mean 0.641 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.0115, ANOVA; Mean Difference (Final Values) = -1.614, 95% CI [-2.851 to -0.378], Standard Error of Mean 0.616 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.9497, ANOVA; Mean Difference (Final Values) = -0.077, 95% CI [-3.047 to 2.893], Standard Error of Mean 1.155 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.5288, ANOVA; Mean Difference (Final Values) = -1.347, 95% CI [-6.467 to 3.773], Standard Error of Mean 1.992 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2595, ANOVA; Mean Difference (Final Values) = -0.296, 95% CI [-0.813 to 0.220], Standard Error of Mean 0.262 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.9605, ANOVA; Mean Difference (Final Values) = -0.013, 95% CI [-0.546 to 0.519], Standard Error of Mean 0.270 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.4107, ANOVA; Mean Difference (Final Values) = -0.207, 95% CI [-0.702 to 0.288], Standard Error of Mean 0.251 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2271, ANOVA; Mean Difference (Final Values) = -0.318, 95% CI [-0.836 to 0.200], Standard Error of Mean 0.263 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9552, ANOVA; Mean Difference (Final Values) = -0.015, 95% CI [-0.535 to 0.506], Standard Error of Mean 0.263 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9899, ANOVA; Mean Difference (Final Values) = -0.003, 95% CI [-0.533 to 0.526], Standard Error of Mean 0.268 — Mean difference (final values) = Least squares mean difference

27. Secondary Outcome: Current Pain During the Hospital Stay Assessed by the Pain NRS
Description: Subject rated scale for average pain intensity over the last 24 hours. Pain was assessed using the question "How much pain do you have right now?" Scores range from 0 (no pain) to 10 (most possible pain).
Time Frame: 4, 8, 12, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, 104, 112, 120, 128, 136, 144, 152, 160, 168, 176, 184, and 192 hours during the hospital stay
Population: MITT. There were not enough subjects with data at 112, 120, 128, 136, 144, 152, 160, 168, 176, 184, and 192 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 87 | 88 | 82
scores on a scale
  4 hours (n=84, 84, 78) | 4.940 (0.345) | 3.554 (0.344) | 4.363 (0.361)
  8 hours (n=82, 79, 75) | 5.083 (0.305) | 4.529 (0.312) | 5.119 (0.323)
  12 hours (n=66, 68, 64) | 4.779 (0.385) | 4.068 (0.375) | 4.784 (0.376)
  24 hours (n=87, 88, 82) | 4.500 (0.265) | 4.545 (0.262) | 4.836 (0.277)
  32 hours (n=79, 78, 69) | 4.450 (0.293) | 4.507 (0.296) | 4.345 (0.315)
  40 hours (n=62, 55, 55) | 3.720 (0.401) | 3.821 (0.412) | 3.902 (0.408)
  48 hours (n=78, 72, 70) | 4.095 (0.276) | 4.069 (0.284) | 3.785 (0.295)
  56 hours (n=62, 56, 57) | 4.015 (0.329) | 3.358 (0.345) | 3.760 (0.343)
  64 hours (n=46, 37, 45) | 4.220 (0.458) | 3.492 (0.480) | 4.578 (0.423)
  72 hours (n=51, 45, 45) | 3.971 (0.344) | 3.271 (0.379) | 3.826 (0.385)
  80 hours (n=19, 24, 24) | 5.312 (0.678) | 2.403 (0.624) | 4.285 (0.691)
  88 hours (n=16, 13, 20) | 4.265 (0.714) | 2.767 (0.803) | 3.914 (0.730)
  96 hours (n=16, 14, 20) | 3.525 (0.729) | 2.532 (0.773) | 2.658 (0.737)
  104 hours (n=7, 3, 7) | 3.501 (0.908) | 2.680 (1.382) | 1.829 (0.972)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 4 hours; Test type: Superiority or Other; p = 0.2211, ANOVA; Mean Difference (Final Values) = 0.578, 95% CI [-0.350 to 1.506], Standard Error of Mean 0.471 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 4 hours; Test type: Superiority or Other; p = 0.0916, ANOVA; Mean Difference (Final Values) = -0.809, 95% CI [-1.750 to 0.132], Standard Error of Mean 0.477 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 8 hours; Test type: Superiority or Other; p = 0.9312, ANOVA; Mean Difference (Final Values) = -0.036, 95% CI [-0.863 to 0.791], Standard Error of Mean 0.420 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 8 hours; Test type: Superiority or Other; p = 0.1658, ANOVA; Mean Difference (Final Values) = -0.591, 95% CI [-1.428 to 0.247], Standard Error of Mean 0.425 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 12 hours; Test type: Superiority or Other; p = 0.9921, ANOVA; Mean Difference (Final Values) = -0.005, 95% CI [-0.958 to 0.948], Standard Error of Mean 0.483 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 12 hours; Test type: Superiority or Other; p = 0.1367, ANOVA; Mean Difference (Final Values) = -0.715, 95% CI [-1.660 to 0.229], Standard Error of Mean 0.479 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.3561, ANOVA; Mean Difference (Final Values) = -0.336, 95% CI [-1.053 to 0.380], Standard Error of Mean 0.364 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.4260, ANOVA; Mean Difference (Final Values) = -0.291, 95% CI [-1.012 to 0.429], Standard Error of Mean 0.366 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 32 hours; Test type: Superiority or Other; p = 0.7975, ANOVA; Mean Difference (Final Values) = 0.105, 95% CI [-0.703 to 0.914], Standard Error of Mean 0.410 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 32 hours; Test type: Superiority or Other; p = 0.6947, ANOVA; Mean Difference (Final Values) = 0.162, 95% CI [-0.650 to 0.974], Standard Error of Mean 0.412 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; 40 hours; Test type: Superiority or Other; p = 0.6954, ANOVA; Mean Difference (Final Values) = -0.182, 95% CI [-1.101 to 0.736], Standard Error of Mean 0.465 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; 40 hours; Test type: Superiority or Other; p = 0.8665, ANOVA; Mean Difference (Final Values) = -0.081, 95% CI [-1.032 to 0.870], Standard Error of Mean 0.481 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.4216, ANOVA; Mean Difference (Final Values) = 0.311, 95% CI [-0.450 to 1.072], Standard Error of Mean 0.386 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.4673, ANOVA; Mean Difference (Final Values) = 0.285, 95% CI [-0.487 to 1.056], Standard Error of Mean 0.391 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; 56 hours; Test type: Superiority or Other; p = 0.5624, ANOVA; Mean Difference (Final Values) = 0.255, 95% CI [-0.614 to 1.125], Standard Error of Mean 0.440 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; 56 hours; Test type: Superiority or Other; p = 0.3705, ANOVA; Mean Difference (Final Values) = -0.402, 95% CI [-1.286 to 0.482], Standard Error of Mean 0.448 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; 64 hours; Test type: Superiority or Other; p = 0.4539, ANOVA; Mean Difference (Final Values) = -0.358, 95% CI [-1.302 to 0.586], Standard Error of Mean 0.476 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; 64 hours; Test type: Superiority or Other; p = 0.0373, ANOVA; Mean Difference (Final Values) = -1.086, 95% CI [-2.107 to -0.065], Standard Error of Mean 0.515 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 19: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.7600, ANOVA; Mean Difference (Final Values) = 0.146, 95% CI [-0.796 to 1.087], Standard Error of Mean 0.476 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 20: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.2506, ANOVA; Mean Difference (Final Values) = -0.555, 95% CI [-1.507 to 0.397], Standard Error of Mean 0.481 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 21: Comparison: Pregabalin (150 mg) vs Placebo; 80 hours; Test type: Superiority or Other; p = 0.2567, ANOVA; Mean Difference (Final Values) = 1.027, 95% CI [-0.770 to 2.823], Standard Error of Mean 0.895 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 22: Comparison: Pregabalin (300 mg) vs Placebo; 80 hours; Test type: Superiority or Other; p = 0.0167, ANOVA; Mean Difference (Final Values) = -1.882, 95% CI [-3.408 to -0.356], Standard Deviation 0.760 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 23: Comparison: Pregabalin (150 mg) vs Placebo; 88 hours; Test type: Superiority or Other; p = 0.6953, ANOVA; Mean Difference (Final Values) = 0.352, 95% CI [-1.456 to 2.159], Standard Error of Mean 0.890 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 24: Comparison: Pregabalin (300 mg) vs Placebo; 88 hours; Test type: Superiority or Other; p = 0.2080, ANOVA; Mean Difference (Final Values) = -1.147, 95% CI [-2.962 to 0.668], Standard Error of Mean 0.894 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 25: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.3805, ANOVA; Mean Difference (Final Values) = 0.867, 95% CI [-1.116 to 2.849], Standard Error of Mean 0.975 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 26: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.8900, ANOVA; Mean Difference (Final Values) = -0.126, 95% CI [-1.965 to 1.713], Standard Error of Mean 0.905 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 27: Comparison: Pregabalin (150 mg) vs Placebo; 104 hours; Test type: Superiority or Other; p = 0.1821, ANOVA; Mean Difference (Final Values) = 1.672, 95% CI [-1.103 to 4.448], Standard Error of Mean 1.080 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 28: Comparison: Pregabalin (300 mg) vs Placebo; 104 hours; Test type: Superiority or Other; p = 0.6505, ANOVA; Mean Difference (Final Values) = 0.851, 95% CI [-3.693 to 5.395], Standard Error of Mean 1.768 — Mean difference (final values) = Least squares mean difference

28. Secondary Outcome: Pain-Related Sleep Interference Post Surgery
Description: The NRS-Sleep: subject rated 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]) rating how pain has interfered with sleep during the past 24 hours. Weekly mean scores were calculated post hospital discharge.
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours 120 hours, 144 hours, 168 hours, and 192 hours post-surgery, Week 2, Week 4, Week 6/ET
Population: MITT. There were not enough subjects with data at 144, 168, and 192 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 86 | 86 | 81
scores on a scale
  24 hours (n=86, 86, 81) | 4.452 (0.359) | 3.671 (0.364) | 5.481 (0.376)
  48 hours (n=82, 82, 77) | 3.830 (0.293) | 3.408 (0.296) | 4.027 (0.309)
  72 hours (n=59, 58, 59) | 2.926 (0.332) | 2.609 (0.349) | 3.645 (0.345)
  96 hours (n=20, 21, 24) | 4.087 (0.539) | 1.645 (0.522) | 3.213 (0.563)
  120 hours (n=6, 4, 7) | 3.194 (1.665) | 7.237 (2.563) | 1.328 (1.598)
  Week 2 (n=80, 73, 71) | 3.837 (0.217) | 4.128 (0.229) | 4.256 (0.239)
  Week 4 (n=76, 65, 67) | 3.181 (0.216) | 3.042 (0.236) | 3.532 (0.241)
  Week 6/ET (n=61, 56, 57) | 2.484 (0.261) | 2.592 (0.265) | 2.748 (0.284)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.0388, ANOVA; Mean Difference (Final Values) = -1.029, 95% CI [-2.004 to -0.053], Standard Error of Mean 0.495 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.0004, ANOVA; Mean Difference (Final Values) = -1.810, 95% CI [-2.798 to -0.822], Standard Error of Mean 0.501 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.6274, ANOVA; Mean Difference (Final Values) = -0.197, 95% CI [-0.995 to 0.601], Standard Error of Mean 0.405 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.1350, ANOVA; Mean Difference (Final Values) = -0.619, 95% CI [-1.432 to 0.194], Standard Error of Mean 0.413 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.1106, ANOVA; Mean Difference (Final Values) = -0.719, 95% CI [-1.605 to 0.166], Standard Error of Mean 0.448 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.0248, ANOVA; Mean Difference (Final Values) = -1.036, 95% CI [-1.939 to -0.133], Standard Error of Mean 0.457 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.2335, ANOVA; Mean Difference (Final Values) = 0.874, 95% CI [-0.582 to 2.330], Standard Error of Mean 0.725 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.0258, ANOVA; Mean Difference (Final Values) = -1.568, 95% CI [-2.939 to -0.198], Standard Error of Mean 0.682 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.3878, ANOVA; Mean Difference (Final Values) = 1.866, 95% CI [-3.207 to 6.939], Standard Error of Mean 1.973 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.1762, ANOVA; Mean Difference (Final Values) = 5.909, 95% CI [-3.740 to 15.559], Standard Error of Mean 3.754 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1754, ANOVA; Mean Difference (Final Values) = -0.515, 95% CI [-1.261 to 0.231], Standard Error of Mean 0.379 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.1413, ANOVA; Mean Difference (Final Values) = -0.569, 95% CI [-1.329 to 0.191], Standard Error of Mean 0.386 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.1731, ANOVA; Mean Difference (Final Values) = -0.419, 95% CI [-1.023 to 0.185], Standard Error of Mean 0.306 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.6829, ANOVA; Mean Difference (Final Values) = -0.128, 95% CI [-0.747 to 0.490], Standard Error of Mean 0.314 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2436, ANOVA; Mean Difference (Final Values) = -0.351, 95% CI [-0.943 to 0.241], Standard Error of Mean 0.300 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1190, ANOVA; Mean Difference (Final Values) = -0.490, 95% CI [-1.108 to 0.127], Standard Error of Mean 0.313 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 17: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.4117, ANOVA; Mean Difference (Final Values) = -0.264, 95% CI [-0.897 to 0.369], Standard Error of Mean 0.321 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 18: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.6294, ANOVA; Mean Difference (Final Values) = -0.156, 95% CI [-0.794 to 0.482], Standard Error of Mean 0.323 — Mean difference (final values) = Least squares mean difference

29. Secondary Outcome: Change From Baseline in Visual Analogue Scale for Anxiety (VAS-Anxiety) Score Prior to Surgery
Description: VAS-Anxiety was administered to measure pre-operative anxiety. Score: 0 = no anxiety to 100 = worst imaginable anxiety.
Time Frame: Day 1, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours prior to surgery
Population: MITT. There were not enough subjects with data at 6 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 83 | 79 | 78
scores on a scale
  Day 1 (n=83, 79, 78) | 6.133 (2.395) | 7.103 (2.450) | 6.992 (2.523)
  1 hour (n=68, 67, 59) | 6.974 (2.787) | 3.272 (2.805) | 6.085 (3.013)
  2 hours (n=75, 76, 63) | 3.792 (2.860) | 6.818 (2.844) | 6.454 (3.126)
  3 hours (n=52, 58, 63) | 7.477 (3.466) | 7.588 (3.188) | 7.313 (3.108)
  4 hours (n=19, 17, 20) | 8.218 (5.803) | 0.109 (6.150) | 10.133 (5.527)
  5 hours (n=3, 4, 8) | 71.190 (16.886) | 29.819 (7.644) | -15.145 (6.572)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Day 1; Test type: Superiority or Other; p = 0.7958, ANOVA; Mean Difference (Final Values) = -0.859, 95% CI [-7.391 to 5.673], Standard Error of Mean 3.315 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Day 1; Test type: Superiority or Other; p = 0.9733, ANOVA; Mean Difference (Final Values) = 0.111, 95% CI [-6.436 to 6.659], Standard Error of Mean 3.322 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 1 hour; Test type: Superiority or Other; p = 0.8220, ANOVA; Mean Difference (Final Values) = 0.889, 95% CI [-6.898 to 8.675], Standard Error of Mean 3.946 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 1 hour; Test type: Superiority or Other; p = 0.4736, ANOVA; Mean Difference (Final Values) = -2.813, 95% CI [-10.542 to 4.917], Standard Error of Mean 3.917 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 2 hours; Test type: Superiority or Other; p = 0.5113, ANOVA; Mean Difference (Final Values) = -2.662, 95% CI [-10.639 to 5.316], Standard Error of Mean 4.045 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 2 hours; Test type: Superiority or Other; p = 0.9266, ANOVA; Mean Difference (Final Values) = 0.365, 95% CI [-7.425 to 8.154], Standard Error of Mean 3.950 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 3 hours; Test type: Superiority or Other; p = 0.9699, ANOVA; Mean Difference (Final Values) = 0.164, 95% CI [-8.423 to 8.751], Standard Error of Mean 4.347 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 3 hours; Test type: Superiority or Other; p = 0.9482, ANOVA; Mean Difference (Final Values) = 0.275, 95% CI [-8.085 to 8.635], Standard Error of Mean 4.232 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 4 hours; Test type: Superiority or Other; p = 0.7969, ANOVA; Mean Difference (Final Values) = -1.915, 95% CI [-16.842 to 13.012], Standard Error of Mean 7.391 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 4 hours; Test type: Superiority or Other; p = 0.1991, ANOVA; Mean Difference (Final Values) = -10.023, 95% CI [-25.533 to 5.487], Standard Error of Mean 7.680 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; 5 hours; Test type: Superiority or Other; p = 0.0321, ANOVA; Mean Difference (Final Values) = 86.335, 95% CI [13.976 to 158.693], Standard Error of Mean 22.737 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; 5 hours; Test type: Superiority or Other; p = 0.0353, ANOVA; Mean Difference (Final Values) = 44.964, 95% CI [5.837 to 84.091], Standard Error of Mean 12.295 — Mean difference (final values) = Least squares mean difference

30. Secondary Outcome: Timed Up-and-Go (TUG)
Description: TUG: time taken in seconds to rise from a standard arm chair, walk to a line on the floor 3 meters away, turn, return and sit down again.
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, Week 2, Week 4, Week 6/ET
Population: MITT. There were not enough subjects with data at 120 (Pregabalin 300 mg only), 144, 168, and 192 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 78 | 71 | 72
seconds
  24 hours (n=45, 47, 46) | 76.153 (10.449) | 79.973 (8.719) | 82.964 (10.174)
  48 hours (n=69, 70, 64) | 80.027 (8.601) | 79.548 (8.111) | 86.842 (8.927)
  72 hours (n=46, 46, 46) | 66.228 (8.429) | 68.373 (8.561) | 80.142 (9.276)
  96 hours (n=14, 14, 22) | 110.780 (45.437) | 43.021 (36.751) | 70.271 (37.742)
  120 hours (n=5, 2, 5) | 52.591 (5.102) | NA (NA) — Value not calculable due to insufficient number of participants reporting results. | 34.078 (4.700)
  Week 2 (n=78, 71, 72) | 22.322 (2.087) | 21.332 (2.091) | 21.678 (2.113)
  Week 4 (n=73, 65, 63) | 18.072 (1.537) | 18.145 (1.527) | 16.535 (1.563)
  Week 6/ET (n=75, 60, 63) | 12.694 (1.226) | 15.140 (1.437) | 13.813 (1.408)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.5736, ANOVA; Mean Difference (Final Values) = -6.812, 95% CI [-30.792 to 17.169], Standard Error of Mean 12.055 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.8003, ANOVA; Mean Difference (Final Values) = -2.991, 95% CI [-26.438 to 20.455], Standard Error of Mean 11.786 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.5125, ANOVA; Mean Difference (Final Values) = -6.815, 95% CI [-27.369 to 13.740], Standard Error of Mean 10.371 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.4773, ANOVA; Mean Difference (Final Values) = -7.294, 95% CI [-27.563 to 12.976], Standard Error of Mean 10.227 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.2142, ANOVA; Mean Difference (Final Values) = -13.915, 95% CI [-36.055 to 8.226], Standard Error of Mean 11.101 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.2989, ANOVA; Mean Difference (Final Values) = -11.769, 95% CI [-34.197 to 10.659], Standard Error of Mean 11.245 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.3829, ANOVA; Mean Difference (Final Values) = 40.510, 95% CI [-53.429 to 134.449], Standard Error of Mean 45.612 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.5531, ANOVA; Mean Difference (Final Values) = -27.250, 95% CI [-120.59 to 66.092], Standard Error of Mean 45.322 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.2738, ANOVA; Mean Difference (Final Values) = 18.513, 95% CI [-89.376 to 126.402], Standard Error of Mean 8.491 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7987, ANOVA; Mean Difference (Final Values) = 0.644, 95% CI [-4.343 to 5.630], Standard Error of Mean 2.519 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8875, ANOVA; Mean Difference (Final Values) = -0.346, 95% CI [-5.177 to 4.485], Standard Error of Mean 2.441 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.4319, ANOVA; Mean Difference (Final Values) = 1.537, 95% CI [-2.324 to 5.398], Standard Error of Mean 1.949 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.4070, ANOVA; Mean Difference (Final Values) = 1.610, 95% CI [-2.223 to 5.443], Standard Error of Mean 1.935 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.4968, ANOVA; Mean Difference (Final Values) = -1.119, 95% CI [-4.371 to 2.133], Standard Error of Mean 1.641 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.4270, ANOVA; Mean Difference (Final Values) = 1.327, 95% CI [-1.972 to 4.626], Standard Error of Mean 1.665 — Mean difference (final values) = Least squares mean difference

31. Secondary Outcome: Range of Motion (ROM) Assessment of the Active Flexion of the Surgical Knee
Description: The degree of active (patient moving the knee) knee flexion and extension tolerated by each subject was recorded. Active ROM in the sitting position was assessed with a goniometer.
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, and 120 hours post surgery, Week 2, Week 4, Week 6/ET
Population: MITT. There were not enough subjects with data at 144, 168, and 192 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 76 | 78 | 69
degrees
  24 hours (n=74, 71, 68) | 54.877 (2.194) | 60.744 (2.248) | 55.738 (2.287)
  48 hours (n=76, 78, 67) | 69.981 (1.984) | 73.370 (1.967) | 69.178 (2.184)
  72 hours (n=52, 52, 50) | 76.516 (2.274) | 79.535 (2.348) | 75.588 (2.406)
  96 hours (n=17, 17, 24) | 78.624 (3.287) | 79.500 (2.936) | 74.194 (2.969)
  120 hours (n=6, 3, 6) | 80.694 (4.890) | 72.694 (7.881) | 81.765 (5.625)
  Week 2 (n=73, 67, 69) | 89.917 (1.589) | 90.332 (1.656) | 87.992 (1.711)
  Week 4 (n=65, 63, 62) | 98.883 (1.870) | 102.237 (1.914) | 96.921 (2.017)
  Week 6/ET (n=67, 54, 63) | 105.352 (1.845) | 106.252 (2.137) | 103.980 (2.051)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.7742, ANOVA; Mean Difference (Final Values) = -0.862, 95% CI [-6.775 to 5.052], Standard Error of Mean 2.999 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.0996, ANOVA; Mean Difference (Final Values) = 5.006, 95% CI [-0.960 to 10.971], Standard Error of Mean 3.025 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.7738, ANOVA; Mean Difference (Final Values) = 0.803, 95% CI [-4.698 to 6.304], Standard Error of Mean 2.790 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.1328, ANOVA; Mean Difference (Final Values) = 4.192, 95% CI [-1.284 to 9.669], Standard Error of Mean 2.778 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.7585, ANOVA; Mean Difference (Final Values) = 0.928, 95% CI [-5.027 to 6.882], Standard Error of Mean 3.012 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.1900, ANOVA; Mean Difference (Final Values) = 3.946, 95% CI [-1.979 to 9.871], Standard Error of Mean 2.997 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.2365, ANOVA; Mean Difference (Final Values) = 4.430, 95% CI [-3.004 to 11.865], Standard Error of Mean 3.693 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.1616, ANOVA; Mean Difference (Final Values) = 5.306, 95% CI [-2.202 to 12.814], Standard Error of Mean 3.730 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.8819, ANOVA; Mean Difference (Final Values) = -1.071, 95% CI [-17.98 to 15.838], Standard Error of Mean 6.911 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.4676, ANOVA; Mean Difference (Final Values) = -9.071, 95% CI [-37.70 to 19.558], Standard Error of Mean 11.700 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.3813, ANOVA; Mean Difference (Final Values) = 1.925, 95% CI [-2.403 to 6.254], Standard Error of Mean 2.195 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2966, ANOVA; Mean Difference (Final Values) = 2.341, 95% CI [-2.070 to 6.751], Standard Error of Mean 2.236 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.4474, ANOVA; Mean Difference (Final Values) = 1.962, 95% CI [-3.122 to 7.046], Standard Error of Mean 2.576 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0416, ANOVA; Mean Difference (Final Values) = 5.316, 95% CI [0.204 to 10.427], Standard Error of Mean 2.590 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.5935, ANOVA; Mean Difference (Final Values) = 1.372, 95% CI [-3.694 to 6.438], Standard Error of Mean 2.566 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.3966, ANOVA; Mean Difference (Final Values) = 2.272, 95% CI [-3.006 to 7.551], Standard Error of Mean 2.674 — Mean difference (final values) = Least squares mean difference

32. Secondary Outcome: ROM Assessment of the Passive Flexion of the Surgical Knee
Description: The degree of passive (movement of the knee with the aid of physical therapist or designee) knee flexion and extension tolerated by each subject was recorded. Passive ROM in the sitting position was assessed with a goniometer.
Time Frame: 24 hours, 48 hours, 72 hours, 96 hours, and 120 hours post surgery, Week 2, Week 4, Week 6/ET
Population: MITT. There were not enough subjects with data at 144, 168, and 192 hours to calculate least squares mean values.
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 85 | 84 | 80
degrees
  24 hours (n=81, 76, 73) | 66.720 (1.990) | 71.523 (2.098) | 64.991 (2.093)
  48 hours (n=78, 80, 70) | 77.714 (1.695) | 81.322 (1.675) | 76.813 (1.809)
  72 hours (n=53, 50, 53) | 84.154 (1.952) | 88.119 (2.041) | 80.984 (1.971)
  96 hours (n=17, 17, 24) | 86.471 (3.553) | 91.460 (3.174) | 80.287 (3.210)
  120 hours (n=5, 3, 6) | 92.160 (1.517) | 97.160 (2.381) | 79.218 (1.682)
  Week 2 (n=79, 71, 73) | 94.767 (1.520) | 96.973 (1.606) | 93.642 (1.647)
  Week 4 (n=72, 62, 65) | 104.548 (1.680) | 107.703 (1.835) | 101.932 (1.851)
  Week 6/ET (n=74, 60, 66) | 110.318 (1.629) | 111.348 (1.884) | 108.944 (1.848)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.5117, ANOVA; Mean Difference (Final Values) = 1.729, 95% CI [-3.457 to 6.916], Standard Error of Mean 2.631 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; 24 hours; Test type: Superiority or Other; p = 0.0154, ANOVA; Mean Difference (Final Values) = 6.532, 95% CI [1.258 to 11.805], Standard Error of Mean 2.675 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.7022, ANOVA; Mean Difference (Final Values) = 0.901, 95% CI [-3.738 to 5.540], Standard Error of Mean 2.353 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; 48 hours; Test type: Superiority or Other; p = 0.0557, ANOVA; Mean Difference (Final Values) = 4.509, 95% CI [-0.110 to 9.129], Standard Error of Mean 2.343 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.2161, ANOVA; Mean Difference (Final Values) = 3.171, 95% CI [-1.874 to 8.215], Standard Error of Mean 2.552 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; 72 hours; Test type: Superiority or Other; p = 0.0058, ANOVA; Mean Difference (Final Values) = 7.135, 95% CI [2.098 to 12.172], Standard Error of Mean 2.548 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.1283, ANOVA; Mean Difference (Final Values) = 6.185, 95% CI [-1.853 to 14.223], Standard Error of Mean 3.993 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; 96 hours; Test type: Superiority or Other; p = 0.0080, ANOVA; Mean Difference (Final Values) = 11.173, 95% CI [3.056 to 19.291], Standard Error of Mean 4.033 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 9: Comparison: Pregabalin (150 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.0018, ANOVA; Mean Difference (Final Values) = 12.941, 95% CI [7.414 to 18.468], Standard Error of Mean 2.150 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 10: Comparison: Pregabalin (300 mg) vs Placebo; 120 hours; Test type: Superiority or Other; p = 0.0038, ANOVA; Mean Difference (Final Values) = 17.941, 95% CI [8.859 to 27.023], Standard Error of Mean 3.533 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 11: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.5953, ANOVA; Mean Difference (Final Values) = 1.125, 95% CI [-3.045 to 5.296], Standard Error of Mean 2.115 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 12: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.1267, ANOVA; Mean Difference (Final Values) = 3.331, 95% CI [-0.952 to 7.613], Standard Error of Mean 2.172 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 13: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2647, ANOVA; Mean Difference (Final Values) = 2.617, 95% CI [-1.997 to 7.231], Standard Error of Mean 2.339 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 14: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.0181, ANOVA; Mean Difference (Final Values) = 5.771, 95% CI [0.995 to 10.548], Standard Error of Mean 2.421 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 15: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.5507, ANOVA; Mean Difference (Final Values) = 1.374, 95% CI [-3.161 to 5.910], Standard Error of Mean 2.299 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 16: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.3164, ANOVA; Mean Difference (Final Values) = 2.404, 95% CI [-2.317 to 7.124], Standard Error of Mean 2.393 — Mean difference (final values) = Least squares mean difference

33. Secondary Outcome: Time From End of Surgery to Meet Hospital Discharge Criteria
Description: The analysis was performed by Kaplan-Meier method with log-rank test.
Time Frame: time from end of surgery up to 192 hours post surgery
Population: MITT
Measure: Mean (Standard Error); unit: hours
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 83 | 84 | 82
hours | 106.802 (6.059) | 112.966 (7.707) | 95.531 (3.385)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Test type: Superiority or Other; p = 0.4365, Log Rank
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Test type: Superiority or Other; p = 0.4023, Log Rank

34. Secondary Outcome: Time From End of Surgery to Actual Discharge
Description: The analysis was performed by Kaplan-Meier method with log-rank test.
Time Frame: time from end of surgery up to 192 hours post surgery
Population: MITT
Measure: Mean (Standard Error); unit: hours
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 78 | 82 | 75
hours | 75.709 (2.798) | 73.906 (2.404) | 78.451 (2.715)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Test type: Superiority or Other; p = 0.4024, Log Rank
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Test type: Superiority or Other; p = 0.1910, Log Rank

35. Secondary Outcome: Satisfaction With Current Pain Medication Measured by the Pain Treatment Satisfaction Scale (PTSS)
Description: Measure of subject satisfaction with treatment for acute or chronic pain. Response range: 1 (strongly agree) to 5 (strongly disagree). Mean scores were calculated and transformed onto a scale of 0-100, range: 0 = worst possible satisfaction to 100 = best possible satisfaction with pain treatment.
Time Frame: Discharge, Week 2, Week 4, Week 6/ET
Population: MITT.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 84 | 84 | 80
scores on a scale
  Discharge (n=84, 84, 80) | 79.897 (1.802) | 80.706 (1.809) | 77.550 (1.890)
  Week 2 (n=22, 20, 18) | 85.274 (4.689) | 85.294 (4.782) | 80.148 (5.201)
  Week 4 (n=30, 27, 19) | 83.608 (3.012) | 84.728 (3.010) | 81.572 (3.765)
  Week 6/ET (n=32, 31, 40) | 74.618 (3.922) | 76.925 (4.187) | 71.962 (4.044)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.3483, ANOVA; Mean Difference (Final Values) = 2.347, 95% CI [-2.573 to 7.268], Standard Error of Mean 2.497 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.2078, ANOVA; Mean Difference (Final Values) = 3.155, 95% CI [-1.766 to 8.077], Standard Error of Mean 2.498 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4299, ANOVA; Mean Difference (Final Values) = 5.126, 95% CI [-7.836 to 18.088], Standard Error of Mean 6.436 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4482, ANOVA; Mean Difference (Final Values) = 5.146, 95% CI [-8.400 to 18.693], Standard Error of Mean 6.726 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6472, ANOVA; Mean Difference (Final Values) = 2.036, 95% CI [-6.818 to 10.890], Standard Error of Mean 4.426 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.4992, ANOVA; Mean Difference (Final Values) = 3.156, 95% CI [-6.129 to 12.442], Standard Error of Mean 4.642 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.6072, ANOVA; Mean Difference (Final Values) = 2.656, 95% CI [-7.578 to 12.891], Standard Error of Mean 5.149 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.3146, ANOVA; Mean Difference (Final Values) = 4.963, 95% CI [-4.789 to 14.714], Standard Error of Mean 4.906 — Mean difference (final values) = Least squares mean difference

36. Secondary Outcome: Satisfaction With Medication Characteristics Measured by the PTSS
Description: as for outcome 35
Time Frame: Discharge, Week 2, Week 4, Week 6/ET
Population: MITT.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 84 | 84 | 80
scores on a scale
  Discharge (n=84, 84, 80) | 85.733 (1.679) | 85.732 (1.685) | 81.556 (1.761)
  Week 2 (n=22, 20, 18) | 91.880 (4.676) | 87.869 (4.769) | 84.583 (5.187)
  Week 4 (n=30, 27, 19) | 88.492 (2.693) | 90.571 (2.691) | 84.323 (3.366)
  Week 6/ET (n=32, 31, 40) | 82.339 (3.729) | 84.571 (3.980) | 76.908 (3.845)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0739, ANOVA; Mean Difference (Final Values) = 4.177, 95% CI [-0.407 to 8.760], Standard Error of Mean 2.326 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0740, ANOVA; Mean Difference (Final Values) = 4.176, 95% CI [-0.409 to 8.761], Standard Error of Mean 2.327 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2615, ANOVA; Mean Difference (Final Values) = 7.298, 95% CI [-5.628 to 20.224], Standard Error of Mean 6.418 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.6266, ANOVA; Mean Difference (Final Values) = 3.286, 95% CI [-10.22 to 16.795], Standard Error of Mean 6.707 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2963, ANOVA; Mean Difference (Final Values) = 4.170, 95% CI [-3.747 to 12.086], Standard Error of Mean 3.958 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1375, ANOVA; Mean Difference (Final Values) = 6.248, 95% CI [-2.054 to 14.550], Standard Error of Mean 4.151 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.2703, ANOVA; Mean Difference (Final Values) = 5.431, 95% CI [-4.298 to 15.161], Standard Error of Mean 4.895 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.1040, ANOVA; Mean Difference (Final Values) = 7.663, 95% CI [-1.607 to 16.933], Standard Error of Mean 4.664 — Mean difference (final values) = Least squares mean difference

37. Secondary Outcome: Satisfaction With Medication Efficacy Measured by the PTSS
Description: as for outcome 35
Time Frame: Discharge, Week 2, Week 4, Week 6/ET
Population: MITT.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 84 | 84 | 80
scores on a scale
  Discharge (n=84, 84, 80) | 74.156 (2.276) | 75.705 (2.284) | 73.577 (2.387)
  Week 2 (n=22, 20, 18) | 78.669 (6.010) | 82.724 (6.129) | 75.713 (6.666)
  Week 4 (n=30, 27, 19) | 78.723 (3.811) | 78.886 (3.808) | 78.823 (4.763)
  Week 6/ET (n=32, 31, 40) | 66.887 (4.958) | 69.367 (5.292) | 67.015 (5.112)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.8545, ANOVA; Mean Difference (Final Values) = 0.579, 95% CI [-5.635 to 6.793], Standard Error of Mean 3.154 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5006, ANOVA; Mean Difference (Final Values) = 2.128, 95% CI [-4.088 to 8.344], Standard Error of Mean 3.155 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7217, ANOVA; Mean Difference (Final Values) = 2.956, 95% CI [-13.66 to 19.569], Standard Error of Mean 8.248 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4203, ANOVA; Mean Difference (Final Values) = 7.011, 95% CI [-10.35 to 24.372], Standard Error of Mean 8.620 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9859, ANOVA; Mean Difference (Final Values) = -0.100, 95% CI [-11.30 to 11.102], Standard Error of Mean 5.600 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9915, ANOVA; Mean Difference (Final Values) = 0.063, 95% CI [-11.68 to 11.811], Standard Error of Mean 5.873 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.9843, ANOVA; Mean Difference (Final Values) = -0.128, 95% CI [-13.06 to 12.808], Standard Error of Mean 6.508 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.7055, ANOVA; Mean Difference (Final Values) = 2.351, 95% CI [-9.974 to 14.677], Standard Error of Mean 6.201 — Mean difference (final values) = Least squares mean difference

38. Secondary Outcome: Overall Satisfaction Measured by the PTSS
Description: as for outcome 35
Time Frame: Discharge, Week 2, Week 4, and Week 6/ET
Population: MITT.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 12 | 17 | 15
scores on a scale
  Discharge (n=12, 17, 15) | 1.845 (0.247) | 1.654 (0.202) | 1.821 (0.219)
  Week 2 (n=6, 4, 4) | 2.333 (0.827) | 1.667 (0.675) | 1.833 (0.893)
  Week 4 (n=4, 3, 4) | 1.149 (0.615) | 2.433 (0.679) | 2.478 (0.629)
  Week 6/ET (n=2, 5, 6) | 1.526 (1.346) | 4.174 (0.784) | 3.878 (0.765)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.9405, ANOVA; Mean Difference (Final Values) = 0.024, 95% CI [-0.614 to 0.661], Standard Error of Mean 0.315 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5641, ANOVA; Mean Difference (Final Values) = -0.167, 95% CI [-0.749 to 0.415], Standard Error of Mean 0.287 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.5226, ANOVA; Mean Difference (Final Values) = 0.500, 95% CI [-1.181 to 2.181], Standard Error of Mean 0.755 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8557, ANOVA; Mean Difference (Final Values) = -0.167, 95% CI [-2.156 to 1.823], Standard Error of Mean 0.893 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1925, ANOVA; Mean Difference (Final Values) = -1.328, 95% CI [-3.596 to 0.940], Standard Error of Mean 0.882 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9654, ANOVA; Mean Difference (Final Values) = -0.045, 95% CI [-2.568 to 2.479], Standard Error of Mean 0.982 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.2350, ANOVA; Mean Difference (Final Values) = -2.352, 95% CI [-6.712 to 2.008], Standard Error of Mean 1.782 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.7420, ANOVA; Mean Difference (Final Values) = 0.296, 95% CI [-1.806 to 2.399], Standard Error of Mean 0.859 — Mean difference (final values) = Least squares mean difference

39. Secondary Outcome: Overall Pain Relief Measured by the PTSS
Description: as for outcome 35
Time Frame: Discharge, Week 2, Week 4, and Week 6/ET
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 12 | 17 | 15
scores on a scale
  Discharge (n=12, 17, 15) | 2.260 (0.258) | 1.696 (0.211) | 2.051 (0.229)
  Week 2 (n=6, 4, 4) | 2.333 (0.827) | 1.667 (0.675) | 1.833 (0.893)
  Week 4 (n=4, 3, 4) | 1.418 (0.713) | 2.612 (0.788) | 2.537 (0.730)
  Week 6/ET (n=2, 5, 6) | 2.067 (1.403) | 4.233 (0.817) | 3.900 (0.797)
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.5299, ANOVA; Mean Difference (Final Values) = 0.208, 95% CI [-0.458 to 0.874], Standard Error of Mean 0.329 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.2442, ANOVA; Mean Difference (Final Values) = -0.355, 95% CI [-0.964 to 0.253], Standard Error of Mean 0.300 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.5226, ANOVA; Mean Difference (Final Values) = 0.500, 95% CI [-1.181 to 2.181], Standard Error of Mean 0.755 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.8557, ANOVA; Mean Difference (Final Values) = -0.167, 95% CI [-2.156 to 1.823], Standard Error of Mean 0.893 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.3240, ANOVA; Mean Difference (Final Values) = -1.119, 95% CI [-3.751 to 1.512], Standard Error of Mean 1.024 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9503, ANOVA; Mean Difference (Final Values) = 0.075, 95% CI [-2.853 to 3.003], Standard Error of Mean 1.139 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.3618, ANOVA; Mean Difference (Final Values) = -1.833, 95% CI [-6.379 to 2.712], Standard Error of Mean 1.858 — Mean difference (final values) = Least squares mean difference
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.7226, ANOVA; Mean Difference (Final Values) = 0.333, 95% CI [-1.859 to 2.525], Standard Error of Mean 0.896 — Mean difference (final values) = Least squares mean difference

40. Secondary Outcome: Number of Subjects With Global Evaluation of Study Medication Scores
Description: The Global Evaluation of Study Medication is a subject-administered single item instrument that records the subject's overall impression (global evaluation) of the study medication by asking the following question: how would you rate the study medication you received for pain? The subject chooses based on a scale of 1 (poor), 2 (fair), 3 (good), or 4 (excellent).
Time Frame: Discharge, Week 2, Week 4, and Week 6/ET
Population: MITT
Measure: Number; unit: participants
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 85 | 84 | 78
participants
  Discharge, Excellent (n=85, 84, 78) | 31 | 27 | 19
  Discharge, Good (n=85, 84, 78) | 31 | 46 | 39
  Discharge, Fair (n=85, 84, 78) | 14 | 6 | 12
  Discharge, Poor (n=85, 84, 78) | 9 | 5 | 8
  Week 2, Excellent (n=22, 20, 18) | 6 | 10 | 5
  Week 2, Good (n=22, 20, 18) | 11 | 4 | 9
  Week 2, Fair (n=22, 20, 18) | 3 | 4 | 1
  Week 2, Poor (n=22, 20, 18) | 2 | 2 | 3
  Week 4, Excellent (n=30, 27, 19) | 13 | 9 | 7
  Week 4, Good (n=30, 27, 19) | 11 | 12 | 8
  Week 4, Fair (n=30, 27, 19) | 4 | 3 | 3
  Week 4, Poor (n=30, 27, 19) | 2 | 3 | 1
  Week 6/ET, Excellent (n=32, 31, 40) | 3 | 7 | 5
  Week 6/ET, Good (n=32, 31, 40) | 17 | 9 | 19
  Week 6/ET, Fair (n=32, 31, 40) | 6 | 5 | 7
  Week 6/ET, Poor (n=32, 31, 40) | 6 | 10 | 9
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.2473, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Discharge; Test type: Superiority or Other; p = 0.0239, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.6118, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Week 2; Test type: Superiority or Other; p = 0.6730, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Pregabalin (150 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.5954, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Pregabalin (300 mg) vs Placebo; Week 4; Test type: Superiority or Other; p = 0.7784, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Pregabalin (150 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.7293, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Pregabalin (300 mg) vs Placebo; Week 6/ET; Test type: Superiority or Other; p = 0.5202, Cochran-Mantel-Haenszel

41. Secondary Outcome: Number of Subjects With Persistent Pain Based on 11-Point Verbal Rating Scale (VRS)
Description: The presence of persistent pain was evaluated on the 11-point VRS. The subject answered the question: how much pain did you experience in the last 24 hours in your operated knee? A zero score of VRS was the only number considered as a "no." Any positive score (1-10) of VRS was consider as "yes."
Time Frame: Month 3, Month 6 (phone call)
Population: MITT
Measure: Number; unit: participants
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 65 | 59 | 61
participants
  Month 3, Yes (n=65, 59, 61) | 22 | 22 | 27
  Month 3, No (n=65, 59, 61) | 43 | 37 | 34
  Month 6, Yes (n=64, 62, 61) | 19 | 15 | 14
  Month 6, No (n=64, 62, 61) | 45 | 47 | 47
Statistical Analysis 1: Comparison: Pregabalin (150 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.1509, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Pregabalin (300 mg) vs Placebo; Month 3; Test type: Superiority or Other; p = 0.3822, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Pregabalin (150 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.2825, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Pregabalin (300 mg) vs Placebo; Month 6; Test type: Superiority or Other; p = 0.7733, Cochran-Mantel-Haenszel

42. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI)
Description: NPSI: subject rated questionnaire to evaluate 5 dimensions of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia). Includes 10 descriptors ranging from 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. Questionnaire generates a score in each relevant dimension. Total score is calculated as the sum of scores of the 10 descriptors, range: 0-100. Higher score indicates greater intensity of pain.
Time Frame: Month 3, Month 6 (phone call)
Population: MITT
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Number analyzed (Participants) | 23 | 24 | 29
scores on a scale
  Burning Spontaneous Pain, Month 3, (n=23, 24, 29) | 1.348 (2.479) | 0.792 (2.085) | 0.828 (1.947)
  Burning Spontaneous Pain, Month 6, (n=22, 15, 15) | 1.091 (2.114) | 1.400 (2.324) | 0.667 (1.113)
  Pressing Spontaneous Pain, Month 3, (n=23, 24, 29) | 1.457 (2.083) | 0.958 (1.574) | 0.948 (1.496)
  Pressing Spontaneous Pain, Month 6, (n=22, 15, 15) | 1.409 (2.158) | 1.333 (1.655) | 0.633 (1.445)
  Paroxysmal Pain, Month 3, (n=23, 24, 29) | 0.804 (1.042) | 1.688 (2.417) | 1.086 (1.909)
  Paroxysmal Pain, Month 6, (n=22, 15, 15) | 1.205 (2.711) | 1.133 (2.175) | 0.533 (1.246)
  Evoked Pain, Month 3, (n=23, 24, 29) | 1.174 (1.700) | 1.319 (2.004) | 0.931 (1.344)
  Evoked Pain, Month 6, (n=22, 15, 15) | 0.636 (0.937) | 1.667 (2.402) | 0.711 (1.298)
  Paresthesia/Dysesthesia, Month 3, (n=23, 24, 29) | 0.848 (1.473) | 0.604 (1.406) | 0.690 (1.160)
  Paresthesia/Dysesthesia, Month 6, (n=22, 15, 15) | 0.773 (1.674) | 0.500 (1.086) | 0.033 (0.129)
  Total Score, Month 3, (n=23, 24, 29) | 0.058 (0.061) | 0.055 (0.075) | 0.045 (0.059)
  Total Score, Month 6, (n=22, 15, 15) | 0.051 (0.074) | 0.061 (0.078) | 0.027 (0.036)

ADVERSE EVENTS:
Arm/Group | Pregabalin (150 mg) | Pregabalin (300 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 11/98 | 11/96 | 5/98
Other Adverse Events (participants affected / at risk) | 76/98 | 76/96 | 81/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (150 mg) (N=98) | Pregabalin (300 mg) (N=96) | Placebo (N=98)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Porcelain gallbladder (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bacterial culture positive (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Muscle flap operation (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Thrombosed varicose vein (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (150 mg) (N=98) | Pregabalin (300 mg) (N=96) | Placebo (N=98)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 9
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 | 3 | 4
Vision blurred (Eye disorders) | 0 | 7 | 0
Constipation (Gastrointestinal disorders) | 24 | 12 | 30
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 5
Nausea (Gastrointestinal disorders) | 29 | 31 | 51
Vomiting (Gastrointestinal disorders) | 14 | 15 | 25
Fatigue (General disorders) | 20 | 15 | 19
Oedema (General disorders) | 1 | 4 | 2
Oedema peripheral (General disorders) | 7 | 9 | 11
Pyrexia (General disorders) | 13 | 16 | 5
Urinary tract infection (Infections and infestations) | 4 | 2 | 4
Anaemia postoperative (Injury, poisoning and procedural complications) | 7 | 7 | 3
Postoperative fever (Injury, poisoning and procedural complications) | 2 | 3 | 4
Procedural nausea (Injury, poisoning and procedural complications) | 5 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 6 | 7 | 5
Body temperature increased (Investigations) | 4 | 5 | 1
Haematocrit decreased (Investigations) | 5 | 4 | 3
Haemoglobin decreased (Investigations) | 6 | 5 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 2 | 6
Disturbance in attention (Nervous system disorders) | 10 | 11 | 11
Dizziness (Nervous system disorders) | 20 | 25 | 16
Headache (Nervous system disorders) | 7 | 3 | 9
Hypoaesthesia (Nervous system disorders) | 3 | 4 | 2
Somnolence (Nervous system disorders) | 24 | 22 | 20
Anxiety (Psychiatric disorders) | 2 | 4 | 6
Confusional state (Psychiatric disorders) | 9 | 10 | 5
Insomnia (Psychiatric disorders) | 8 | 12 | 17
Dysuria (Renal and urinary disorders) | 5 | 4 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 12 | 21
Hypertension (Vascular disorders) | 4 | 3 | 7
Hypotension (Vascular disorders) | 12 | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.